## 1.0 Title Page

## **Statistical Analysis Plan**

## Study M15-554

A Phase 3, Randomized, Double-Blind, Study Comparing Upadacitinib (ABT-494) to Placebo in Subjects with Active Psoriatic Arthritis Who Have a History of Inadequate Response to at Least One Biologic Disease Modifying Anti-Rheumatic Drug (bDMARD) – SELECT – PsA 2

Date: 24 May 2021

Version 3.0

| 7 |
|------------------------------------------|
| 10G |
| es/ |
| 7 |
| 7 |
| 10 |
| 10 |
| 10 |
| dows10 |
| 10 |
| 11 |
| s, Medical<br>edications <mark>16</mark> |
| 16 |
| 19 |
| 19 |
| 20 |
| <mark>20</mark> |
| 22 |
| 22 |
| 24 |
| 24 |
| 24 |
| ly24 |
| ts25 |
| 27 |
| cy Endpoint27 |
| Endpoint28 |
| 28 |
| 32 |

| 9.2.5 | Handling of Multiplicity |
|---|---|
| 9.2.6 | Efficacy Subgroup Analysis |
| 9.3 | Long-Term Efficacy Analysis |
| 9.4 | Efficacy Variables Definitions and Conventions39 |
| 9.4.1 | ACR Criteria |
| 9.4.2 | Joint Evaluation |
| 9.4.3 | Patient's Global Assessment of Disease Activity Numeric Rating Scale (NRS)44 |
| 9.4.4 | Physician's Global Assessment of Disease Activity Numeric Rating Scale (NRS)44 |
| 9.4.5 | Patient's Assessment of Pain Numeric Rating Sale (NRS)44 |
| 9.4.6 | Disease Activity Score (DAS28)44 |
| 9.4.7 | Disease Activity in Psoriatic Arthritis (DAPSA) Score45 |
| 9.4.8 | PsA Disease Activity Score (PASDAS)46 |
| 9.4.9 | Disability Index of Health Assessment Questionnaire (HAQ-DI)47 |
| 9.4.10 | Static Investigator Global Assessment of Psoriasis (sIGA)47 |
| 9.4.11 | Psoriasis Area Severity Index (PASI) |
| 9.4.12 | Minimum Disease Activity for PsA |
| 9.4.13 | Self-Assessment of Psoriasis Symptoms (SAPS)50 |
| 9.4.14 | Leeds Dactylitis Index (LDI) and Dactylitis Count50 |
| 9.4.15 | Leeds and SPARCC Enthesitis Indices and Total Enthesitis Count51 |
| 9.4.16 | Body Surface Area (BSA) – Psoriasis |
| 9.4.17 | Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and Morning Stiffness Score |
| 9.4.18 | Modified Psoriatic Arthritis Response Criteria (PsARC)53 |
| 9.4.19 | Ankylosing Spondylitis Disease Activity Score (ASDAS)54 |
| 9.4.20 | FACIT-Fatigue Questionnaire (FACIT-F)55 |
| 9.4.21 | EuroQoL-5D (EQ-5D-5L)55 |
| 9.4.22 | Form SF-36v2 |
| 9.4.23 | Work Productivity and Activity Impairment Questionnaire Psoriatic Arthritis (WPAI) |
| 9.4.24 | Health Resource Utilization (HRU) Questionnaire |
| 10.0 | Safety Analysis59 |

| 10.1 General Considerations 59 10.2 Analysis of Adverse Events 61 10.2.1 Analysis of Adverse Events Prior to Protocol-Defined Treatment Switching 62 10.2.1.1 Adverse Events Overview 62 10.2.1.2 Adverse Events by System Organ Class and Preferred Term 62 10.2.1.3 TEAEs by Maximum Severity 63 10.2.1.4 TEAEs by Relationship 63 10.2.1.5 Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term 63 10.2.1.6 Adverse Events of Special Interest 64 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure 67 10.2.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.3 Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.3.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation 69 10.3.1 Variables and Units 69 < | | | |
|---|---|---|---|
| 10.2.1 Analysis of Adverse Events Prior to Protocol-Defined Treatment Switching 62 10.2.1.1 Adverse Events Overview 62 10.2.1.2 Adverse Events by System Organ Class and Preferred Term 62 10.2.1.3 TEAEs by Maximum Severity 63 10.2.1.4 TEAEs by Relationship 63 10.2.1.5 Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term 63 10.2.1.6 Adverse Events of Special Interest 64 10.2.2 Analysis of Long-Term Adverse Event Rates 67 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure 67 10.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.3 Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation 69 10.3 Analysis of Laboratory Data 69 10.3.1 Variables and Units 69 10.3.2 Analysis of Laboratory Data Through Week 24 71 10.3.2.2 Asses | 10.1 | General Considerations | 59 |
| Switching 62 10.2.1.1 Adverse Events Overview 62 10.2.1.2 Adverse Events by System Organ Class and Preferred Term 62 10.2.1.3 TEAEs by Maximum Severity 63 10.2.1.4 TEAEs by Relationship 63 10.2.1.5 Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term 63 10.2.1.6 Adverse Events of Special Interest 64 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure 67 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.3 Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation 69 10.3 Analysis of Laboratory Data 69 10.3.1 Variables and Units 69 10.3.2.1 Assessment of Shift from Baseline in Clinical Laboratory Variables | 10.2 | Analysis of Adverse Events | 61 |
| 10.2.1.1 Adverse Events Overview | 10.2.1 | Analysis of Adverse Events Prior to Protocol-Defined Treatment | |
| 10.2.1.2 Adverse Events by System Organ Class and Preferred Term | | | |
| 10.2.1.3 TEAEs by Maximum Severity 63 10.2.1.4 TEAEs by Relationship 63 10.2.1.5 Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term 63 10.2.1.6 Adverse Events of Special Interest 64 10.2.2 Analysis of Long-Term Adverse Event Rates 67 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure 67 10.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.3 Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation 69 10.3 Analysis of Laboratory Data 69 10.3.1 Variables and Units 69 10.3.2 Analysis of Laboratory Data Through Week 24 71 10.3.2.1 Assessment of Clinical Laboratory Variables 71 10.3.2.3 Assessment of Potentially Clinical Significant Laboratory Values 72 10.3.3.4 Assessment of Clinical Laboratory Variables 73 10.3.3.1 Ass | 10.2.1.1 | Adverse Events Overview | 62 |
| 10.2.1.4 TEAEs by Relationship | 10.2.1.2 | Adverse Events by System Organ Class and Preferred Term | 62 |
| 10.2.1.5 Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term | 10.2.1.3 | TEAEs by Maximum Severity | 63 |
| Related Adverse Events by System Organ Class and Preferred Term | 10.2.1.4 | TEAEs by Relationship | 63 |
| Term 63 10.2.1.6 Adverse Events of Special Interest 64 10.2.2 Analysis of Long-Term Adverse Event Rates 67 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure 67 10.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.3 Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation 69 10.3 Analysis of Laboratory Data 69 10.3.1 Variables and Units 69 10.3.2 Analysis of Laboratory Data Through Week 24 71 10.3.2.1 Assessment of Clinical Laboratory Variables 71 10.3.2.2 Assessment of Potentially Clinical Significant Laboratory Values 72 10.3.2.3 Assessment of Liver Elevations 72 10.3.3.1 Assessment of Clinical Laboratory Variables 73 10.3.3.2 Assessment of Potentially Clinical Significant Laboratory Values 74 10.3.3.3 Assessment o | 10.2.1.5 | 1 , , , | |
| 10.2.2 Analysis of Long-Term Adverse Event Rates 67 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure 67 10.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.3 Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT 68 10.2.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation 69 10.3 Analysis of Laboratory Data 69 10.3.1 Variables and Units 69 10.3.2 Analysis of Laboratory Data Through Week 24 71 10.3.2.1 Assessment of Clinical Laboratory Variables 71 10.3.2.2 Assessment of Shift from Baseline in Clinical Laboratory Variables 72 10.3.2.3 Assessment of Potentially Clinical Significant Laboratory Values 72 10.3.3 Analysis of Long-Term Laboratory Data 73 10.3.3.1 Assessment of Clinical Laboratory Variables 73 10.3.3.2 Assessment of Potentially Clinical Significant Laboratory Values 74 10.3.3.3 Assessment of Potentially Clinical Significant Laboratory Values 74 < | | Term | 63 |
| 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure | 10.2.1.6 | Adverse Events of Special Interest | 64 |
| Study Drug Exposure | 10.2.2 | Analysis of Long-Term Adverse Event Rates | 67 |
| Exposure by SOC and PT | 10.2.2.1 | • | 67 |
| Study Drug Exposure by SOC and PT | 10.2.2.2 | <u>.</u> | 68 |
| Adverse Events Leading to Study Drug Discontinuation 69 10.3 Analysis of Laboratory Data 69 10.3.1 Variables and Units 69 10.3.2 Analysis of Laboratory Data Through Week 24 71 10.3.2.1 Assessment of Clinical Laboratory Variables 71 10.3.2.2 Assessment of Shift from Baseline in Clinical Laboratory Variables 71 10.3.2.3 Assessment of Potentially Clinical Significant Laboratory Values 72 10.3.2.4 Assessment of Liver Elevations 72 10.3.3 Analysis of Long-Term Laboratory Data 73 10.3.3.1 Assessment of Clinical Laboratory Variables 73 10.3.3.2 Assessment of Potentially Clinical Significant Laboratory Values 74 10.3.3.3 Assessment of Potentially Clinical Significant Laboratory Values 74 10.3.3.3 Assessment of Liver Elevations 75 | 10.2.2.3 | <u> </u> | 68 |
| 10.3.1Variables and Units6910.3.2Analysis of Laboratory Data Through Week 247110.3.2.1Assessment of Clinical Laboratory Variables7110.3.2.2Assessment of Shift from Baseline in Clinical Laboratory<br>Variables7110.3.2.3Assessment of Potentially Clinical Significant Laboratory Values7210.3.2.4Assessment of Liver Elevations7210.3.3Analysis of Long-Term Laboratory Data7310.3.3.1Assessment of Clinical Laboratory Variables7310.3.3.2Assessment of Potentially Clinical Significant Laboratory Values7410.3.3.3Assessment of Liver Elevations75 | 10.2.2.4 | ` | 69 |
| 10.3.2 Analysis of Laboratory Data Through Week 24 | 10.3 | Analysis of Laboratory Data | 69 |
| 10.3.2.1 Assessment of Clinical Laboratory Variables 71 10.3.2.2 Assessment of Shift from Baseline in Clinical Laboratory Variables 71 10.3.2.3 Assessment of Potentially Clinical Significant Laboratory Values 72 10.3.2.4 Assessment of Liver Elevations 72 10.3.3 Analysis of Long-Term Laboratory Data 73 10.3.3.1 Assessment of Clinical Laboratory Variables 73 10.3.3.2 Assessment of Potentially Clinical Significant Laboratory Values 74 10.3.3.3 Assessment of Liver Elevations 75 | 10.3.1 | Variables and Units | 69 |
| 10.3.2.2 Assessment of Shift from Baseline in Clinical Laboratory Variables | 10.3.2 | Analysis of Laboratory Data Through Week 24 | 71 |
| Variables | 10.3.2.1 | Assessment of Clinical Laboratory Variables | 71 |
| 10.3.2.4Assessment of Liver Elevations7210.3.3Analysis of Long-Term Laboratory Data7310.3.3.1Assessment of Clinical Laboratory Variables7310.3.3.2Assessment of Potentially Clinical Significant Laboratory Values7410.3.3.3Assessment of Liver Elevations75 | 10.3.2.2 | | 71 |
| 10.3.2.4Assessment of Liver Elevations7210.3.3Analysis of Long-Term Laboratory Data7310.3.3.1Assessment of Clinical Laboratory Variables7310.3.3.2Assessment of Potentially Clinical Significant Laboratory Values7410.3.3.3Assessment of Liver Elevations75 | 10.3.2.3 | Assessment of Potentially Clinical Significant Laboratory Values | 72 |
| 10.3.3.1 Assessment of Clinical Laboratory Variables | 10.3.2.4 | | |
| 10.3.3.1 Assessment of Clinical Laboratory Variables | 10.3.3 | Analysis of Long-Term Laboratory Data | 73 |
| 10.3.3.2 Assessment of Potentially Clinical Significant Laboratory Values74 10.3.3.3 Assessment of Liver Elevations | 10.3.3.1 | · | |
| 10.3.3.3 Assessment of Liver Elevations | 10.3.3.2 | • | |
| | 10.4 | Analysis of Vital Signs | 75 |

| 10.4.1 | Variables and Criteria Defining Abnormality | 75 |
|---|---|---|
| 10.4.2 | Analysis of Vital Signs Through Week 24 | |
| 10.4.3 | Analysis of Long-Term Vital Signs | |
| 11.0 | Summary of Changes | |
| 11.1 | Summary of Changes between the Previous Version and the | •••• |
| 11.1 | Current Version | 77 |
| 12.0 | Version History | 79 |
| 13.0 | References | |
| List of Ta | ables | |
| Table 1. | Analysis Windows for Efficacy Analysis for Period 1 (for ACR Components, TJC28, SJC28, ESR and Derived Endpoints <sup>a</sup> ) and Safety Analysis for Period 1 (for Lab Values [Clinical Chemistry, Hematology, Urinalysis] and Vital Signs/Weight) | 13 |
| Table 2. | Analysis Windows for Efficacy Analysis for Period 1 (for SF-36, EQ-5D-5L, FACIT-F, WPAI, BASDAI, HRU and Derived Endpoints <sup>a</sup> ) | 14 |
| Table 3. | Analysis Windows for Safety Analysis for Period 1 (for Total Cholesterol, HDL-C, LDL-C, Triglycerides, Advanced Lipid Testing <sup>a</sup> ) | |
| Table 4. | Analysis Windows for Efficacy Analysis for Period 1 (for BSA-Psoriasis, PASI, sIGA, LDI, LEI, SPARCC Enthesitis Index and Derived Endpoints <sup>a</sup> ) | 15 |
| Table 5. | Analysis Windows for Efficacy Analysis for Period 1 (for SAPS) | 15 |
| Table 6. | Subgroups for Efficacy Analysis | 37 |
| Table 7. | Anatomical Joints Assessed for Calculation of Tender and Swollen Joint Counts (TJC68 and SJC66) | 43 |
| Table 8. | Anatomical Joints for DAS28 (CRP) Calculation | 45 |
| Table 9. | AESI for Upadacitinib with SMQs/CMQs/PTs Searches | 65 |
| Table 10. | List of Laboratory Variables | 69 |
| Table 11. | Criteria for Potentially Clinically Significant Vital Sign Findings | 76 |
| Table 12. | SAP Version History Summary | 79 |



## **List of Figures** Study Design ......9 Figure 1. Figure 2. Graphical Multiple Testing Procedure......36 **List of Appendices** Appendix A. SAS Procedure for Mantel-Haenszel Test ......80 Appendix B. Tipping Point Analysis for ACR20 at Week 12 ......81 Appendix C. Tipping Point Analysis for Key Secondary Continuous Endpoint .........82 Appendix D. Exposure Adjusted AE Rate Difference and Normal Approximation Based 95% Confidence Interval (Liu, F et al. 2006<sup>5</sup>)......85 Statistical Analysis to Account for the Impact of COVID-19 Appendix E. Pandemic 86



## 3.0 Introduction

This statistical analysis plan (SAP) describes the statistical analyses to be completed by the Data and Statistical Science Department for upadacitinib Study M15-554. It provides details to further elaborate statistical methods as outlined in the protocol.

Pharmacokinetic and biomarker analyses will be performed separately and are not in the scope of this SAP.

Unless noted otherwise, all analyses will be performed using SAS version 9.2 or later (SAS Institute Inc., Cary, NC 27513) under the UNIX operating system.

## 4.0 Study Objectives, Design and Procedures

## 4.1 Study Objectives

#### Period 1

To compare the efficacy of upadacitinib 15 mg once daily (QD) and 30 mg QD versus placebo for the treatment of signs and symptoms in subjects with moderately to severely active Psoriatic Arthritis (PsA) who have an inadequate response to biologic DMARDs (Bio-IR).

To compare the safety and tolerability of upadacitinib 15 mg QD and 30 mg QD versus placebo in subjects with moderately to severely active PsA who have an inadequate response to biologic DMARDs.

#### Period 2

To evaluate the long-term safety, tolerability and efficacy of upadacitinib 15 mg QD and 30 mg QD in subjects with PsA who have completed Period 1.

## 4.2 Overall Study Design and Plan

This is a Phase 3 multicenter study that includes two periods. Period 1 is 56 weeks in duration and includes a 24-week randomized, double-blind, parallel-group, placebo-

controlled period followed by an additional 32 weeks of blinded active treatment (Weeks 24 – 56). Period 1 is designed to compare the safety, tolerability, and efficacy of upadacitinib 15 mg QD and 30 mg QD versus placebo in subjects with moderately to severely active PsA who have an inadequate response to bDMARDs (Bio-IR). Period 2 is an open-label (blinded until the last subject completes the last visit of Period 1), long-term extension of up to a total treatment duration of approximately 3 years to evaluate the safety, tolerability and efficacy of upadacitinib 15 mg QD and 30 mg QD in subjects with PsA who have completed Period 1. In certain countries (Belgium, Czech Republic, France, Greece, Hungary, Japan, New Zealand, and Portugal), subjects will continue to receive upadacitinib therapy after Week 152 until regulatory approval and/or applicable local reimbursement approval of the study drug in the respective country. Starting with Amendment 7.01.01, subjects in Japan receiving upadacitinib 30 mg QD will be switched to upadacitinib 15 mg QD. For other countries, starting with Amendment 8 and 8.01, subjects receiving upadacitinib 30 mg QD will be switched to upadacitinib 15 mg QD.

The study is designed to enroll approximately 630 subjects at approximately 165 study centers worldwide to meet scientific and regulatory objectives without enrolling an undue number of subjects in alignment with ethical considerations.

Subjects who meet eligibility criteria will be randomized in a 2:2:1:1 ratio using an Interactive Response Technology (IRT) to receive double-blind study drug in one of the following treatment groups:

- Group 1: Upadacitinib 15 mg QD, N = 210)
- Group 2: Upadacitinib 30 mg QD, N = 210)
- Group 3: Placebo, N = 105 (Day 1 to Week 24) → Upadacitinib 15 mg QD (Week 24 and thereafter)
- Group 4: Placebo, N = 105 (Day 1 to Week 24) → Upadacitinib 30 mg QD (Week 24 and thereafter)

Randomization will be stratified by extent of psoriasis ( $\geq 3\%$  body surface area [BSA] or < 3% BSA), current use of at least 1 DMARD (Yes or No), and number of prior failed

biologic DMARDs (1 vs > 1), except for subjects from Japan, for which randomization will be stratified by extent of psoriasis ( $\geq$  3% body surface area [BSA] or < 3% BSA) only.

A schematic of the overall study design is shown in Figure 1 below. For a more detailed description of the study design, refer to Section 5.0 of the most up-to-date version of the study protocol.

Figure 1. Study Design



- a. At Week 16 rescue therapy will be offered to subjects classified as non-responders (defined as not achieving at least 20% improvement in either or both tender joint count (TJC) and swollen joint count (SJC) at both Week 12 and Week 16) as described in Section 5.2.3.4 of the most up-to-date version of the study protocol.
- b. At Week 24, all placebo subjects will switch to upadacitinib 15 mg QD or 30 mg QD (1:1 ratio) regardless of response.
- c. Refer to details above in Protocol amendment 8/later version Section 5.1 regarding completion of the study after Week 152.

Note: For subjects in Japan only: Upon approval of protocol amendment 7.01.01, subjects receiving upadacitinib 30 mg QD will be switched to upadacitinib 15 mg QD prior to marketing approval in Japan for the treatment of psoriatic arthritis.

Note: Upon approval of protocol amendment 8 and 8.01, subjects receiving upadacitinib 30 mg QD will be switched to upadacitinib 15 mg QD at their next scheduled study visit in other countries.



## 4.3 Sample Size

The planned total sample size of 630 for this study provides at least 90% power for a 20% difference in ACR20 response rate (assuming a placebo ACR20 response rate of 20%). It will also provide at least 90% power for the majority of the key secondary endpoints. All power and sample size calculations are performed at a two-sided significance level of 0.025 and accounting for a 10% dropout rate.

## 4.4 Week 24 Analysis and Data Base Lock

After the last subject completes the Week 24 study visit, an unblinded analysis will be conducted for the purpose of initial regulatory submission. To maintain integrity of the trial during the blinded 56-week period (Period 1), study sites and subjects will remain blinded until all subjects have reached Week 56.

## 4.5 Data Monitoring Committee (DMC) Activities

An independent external Data Monitoring Committee (DMC) is used to review unblinded safety data at regular intervals during the conduct of the study. The DMC will provide recommendation to an AbbVie Point of Contact on whether to continue, modify, or terminate studies after each review. When needed, high-level unblinded efficacy data may also be requested by the DMC and be reviewed so that the DMC can assess benefit:risk of any emerging safety differences.

## 5.0 Analysis Populations and Analysis Windows

## 5.1 Analysis Populations

## **Full Analysis Set (FAS)**

The Full Analysis Set (FAS) includes all randomized subjects who received at least one dose of study drug. The FAS will be used for all efficacy and baseline analyses.



#### Per Protocol Analysis Set

The Per Protocol Analysis Set represents a subset of the FAS and consists of all FAS subjects who did not have any major protocol deviations that are determined to have a potential impact on the primary efficacy endpoint up to Week 12 in Period 1 of the study. Additional analysis of the primary efficacy endpoint will be conducted on the Per Protocol analysis set, in order to evaluate the impact of protocol deviations.

Protocol deviations with potential to affect the primary efficacy endpoint (key ICH deviations and other clinically significant non-ICH deviations) will be identified prior to the Week 24 database lock.

#### Safety Analysis Set

The Safety Analysis Set consists of all subjects who received at least one dose of study drug. For the Safety Analysis Set, subjects will be analyzed "as treated," regardless of the treatment randomized. "As treated" is determined by the treatment the subject received during the majority of the subject's drug exposure time in the analysis period.

## 5.2 Analysis Windows

#### **Definition of Study Days (Days Relative to the First Dose of Study Drug)**

Study Days are calculated for each collection date relative to the date of the first dose of study drug. It is defined as the number of days between the date of the first dose of study drug and the collection date. Study days are negative values when the collection date of interest is prior to the first study drug dose date. Study days are positive values when the collection date of interest is on or after the first study drug dose date. The day of the first dose of study drug is defined as Study Day 1, while the day prior to the first study drug dose is defined as Study Day –1 (there is no Study Day 0). Study days are used to map actual study visits to the protocol-specified study visits.



#### **Definition of Analysis Windows**

The following rules will be applied to assign actual subject visits to protocol-specified visits. For each protocol-specified study visit, a target study day will be identified to represent the corresponding visit along with a window around the target day. Windows will be selected in a non-overlapping fashion so that a collection date does not fall into multiple visit windows. If a subject has two or more actual visits in one visit window, the visit closest to the target day will be used for analysis. If two visits are equidistant from the target day, then the later visit will be used for analysis.

The visit window and the target study day for each protocol-specified visit in Period 1 are displayed in Table 1, Table 2, Table 3, Table 4, and Table 5 (depending on the different visit schedules of different endpoints). Visit windows for protocol-specified visits in Period 2 are defined similarly.



Table 1. Analysis Windows for Efficacy Analysis for Period 1 (for ACR Components, TJC28, SJC28, ESR and Derived Endpoints<sup>a</sup>) and Safety Analysis for Period 1 (for Lab Values [Clinical Chemistry, Hematology, Urinalysis] and Vital Signs/Weight)

| Protocol Specified<br>Visit Week | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | -99 | 1 <sup>b</sup> | 1 |
| 2 | 2 | 15 | 22 |
| 4 | 23 | 29 | 43 |
| 8 | 44 | 57 | 71 |
| 12 | 72 | 85 | 99 |
| 16 | 100 | 113 | 127 |
| 20 | 128 | 141 | 155 |
| 24 | 156 | 169 | Min (183, first dose date from Week 24 dispensed kit) |
| 28 | Min (183, first dose date from Week 24 dispensed kit) + 1 | 197 | 211 |
| 32 | 212 | 225 | 239 |
| 36 | 240 | 253 | 281 |
| 44 | 282 | 309 | 351 |
| 56 | 352 | 393 | 435 |

a. ACR20/50/70 response rates, DAS28 (CRP), DAS28 (ESR), PsARC, DAPSA, proportion of subjects achieving a clinically meaningful improvement in HAQ-DI (≥ 0.35).

b. Day of first dose of study drug.



Table 2. Analysis Windows for Efficacy Analysis for Period 1 (for SF-36, EQ-5D-5L, FACIT-F, WPAI, BASDAI, HRU and Derived Endpoints<sup>a</sup>)

| Protocol Specified<br>Visit Week | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | <b>–99</b> | 1 <sup>b</sup> | 1 |
| 12 | 2 | 85 | 127 |
| 24 | 128 | 169 | Min (211, first dose date from Week 24 dispensed kit) |
| 36 | Min (211, first dose date from<br>Week 24 dispensed kit) + 1 | 253 | 323 |
| 56 | 324 | 393 | 435 |

a. PASDAS, BASDAI 50 response rates, Change from baseline in Morning stiffness (mean of BASDAI Questions 5 and 6), ASDAS, proportion of subjects with ASDAS Inactive Disease, proportion of subjects with ASDAS Major Improvement, proportion of subjects with ASDAS Clinically Important Improvement.

Table 3. Analysis Windows for Safety Analysis for Period 1 (for Total Cholesterol, HDL-C, LDL-C, Triglycerides, Advanced Lipid Testing<sup>a</sup>)

| Protocol Specified<br>Visit Week | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | -99 | 1 <sup>b</sup> | 1 |
| 4 | 2 | 29 | 57 |
| 12 | 58 | 85 | 127 |
| 24 | 128 | 169 | Min (211, first dose date from Week 24 dispensed kit) |

a. Advanced lipid testing is exploratory and may not be performed and/or be reported in the CSR.

b. Day of first dose of study drug.

b. Day of first dose of study drug.

Table 4. Analysis Windows for Efficacy Analysis for Period 1 (for BSA-Psoriasis, PASI, sIGA, LDI, LEI, SPARCC Enthesitis Index and Derived Endpoints<sup>a</sup>)

| Protocol Specified<br>Visit Week | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | -99 | 1 <sup>b</sup> | 1 |
| 12 | 2 | 85 | 99 |
| 16 | 100 | 113 | 141 |
| 24 | 142 | 169 | Min (211, first dose date from Week 24 dispensed kit) |
| 36 | Min (211, first dose date from Week 24 dispensed kit) + 1 | 253 | 323 |
| 56 | 324 | 393 | 435 |

a. MDA, dactylitis count/total enthesitis count, proportion of subjects with resolution of dactylitis/enthesitis (out of all sites, or the sites included in SPARCC or LEI), PAISI75/90/100, proportion of subjects achieving a static Investigator Global Assessment of psoriasis (sIGA) score of 0 or 1 and at least a 2-point improvement from baseline.

Table 5. Analysis Windows for Efficacy Analysis for Period 1 (for SAPS)

| Protocol Specified<br>Visit Week | Lower Bound | Target Day | Upper Bound |
|---|---|---|---|
| Baseline | <b>-99</b> | 1ª | 1 |
| 16 | 2 | 113 | 141 |
| 24 | 142 | 169 | Min (211, first dose date from Week 24 dispensed kit) |
| 36 | Min (211, first dose date from<br>Week 24 dispensed kit) + 1 | 253 | 323 |
| 56 | 324 | 393 | 435 |

a. Day of first dose of study drug.

b. Day of first dose of study drug.



## 6.0 Demographics, Baseline Characteristics, Medical History, and Previous/Concomitant Medications

## 6.1 Demographics and Baseline Characteristics

Demographic and baseline characteristics information will be collected at the Baseline visit of the study and will be summarized for the FAS. The number of observations, mean, standard deviation, median, minimum and maximum will be summarized for continuous variables. Categorical or discrete variables will be summarized via frequencies and percentages. Summary statistics will be computed for each treatment group and overall.

#### Main Demographic and Baseline Characteristics

- Sex (male, female)
- Age (years)
- Age Categories ( $< 65, 65 < 75, \ge 75 \text{ years}$ )
- Race (White, Black or African American, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, Asian, Other)
- Geographic Region (North America, Western Europe and Oceania, Eastern Europe, Latin-America, Asia, and Other)
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino)
- Weight (kg)
- Height (cm)
- Body Mass Index (BMI) (kg/m<sup>2</sup>)
- Body Mass Index (BMI) Category (kg/m<sup>2</sup>) (BMI  $\leq$  25, BMI  $\geq$  25)

## **PsA Medical History, Prior and Baseline Treatments**

- Duration of PsA symptoms in years
- Duration of PsA diagnosis in years
- Rheumatoid Factor (RF) status: Positive or Negative

- Anti-CCP status: Positive or Negative
- Number of prior non-biologic DMARDs  $(0, 1, 2, \ge 3)$
- Number of prior biologic DMARDs  $(0, 1, 2, \ge 3)$
- Number of prior biologic DMARDs other than anti-TNF  $(0, 1, 2, \ge 3)$
- Number of prior anti-TNFs  $(0, 1, 2, \ge 3)$
- Number of prior failed biologic DMARDs  $(0, 1, 2, \ge 3)$
- Current use of at least 1 non-biologic DMARD at baseline (Yes or No)
- Current NSAID use at baseline (Yes or No)
- Current Corticosteroid use at baseline (Yes or No)
- Concomitant non-biologic DMARD at baseline (MTX alone, MTX and other non-biologic DMARD, non-biologic DMARD other than MTX)

#### **Baseline Disease Characteristics**

- Tender joint count (TJC68) defined as the number of tender joints out of 68 assessed joints
- Swollen joint count (SJC66) defined as the number of swollen joints out of 66 assessed joints
- Physician's global assessment of Disease Activity Numeric Rating Scale (0 - 10 NRS)
- Patient's assessment of pain (0 10 NRS)
- Patient's assessment of disease activity (0 10 NRS)
- Health Assessment Questionnaire Disability Index (HAQ-DI)
- High sensitivity C-reactive protein (hsCRP)
- Categories for hsCRP: equal or below vs. above ULN (2.87 mg/L)
- Body Surface Area (BSA) with Psoriasis (as categorical with  $< 3\%, \ge 3\%$ )
- Body Surface Area (BSA) with Psoriasis (as continuous for subjects with BSA-Ps > 0%)
- Static Investigator Global Assessment of Psoriasis (sIGA) (as a categorical variable)



- Psoriasis Area and Severity Index (PASI) score (for subjects with ≥ 3% Body Surface Area (BSA) psoriasis)
- Erythrocyte sedimentation rate (ESR)
- Psoriatic arthritis disease activity score (PASDAS)
- Disease Activity In Psoriatic Arthritis (DAPSA) score
- Presence of Dactylitis (defined as LDI > 0)
- Leeds Dactylitis Index (LDI) (out of subjects with presence of dactylitis (LDI > 0))
- Total dactylitis count (out of subjects with presence of dactylitis (LDI > 0))
- Presence of Enthesitis (defined as total enthesitis count > 0)
- Total enthesitis count (out of subjects with presence of enthesitis (total enthesitis count > 0))
- Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index (out of subjects with SPARCC Enthesitis Index > 0)
- Leeds Enthesitis Index (LEI) (out of subjects with LEI > 0)
- DAS28 [CRP]
- DAS28 [ESR]
- Presence of Psoriatic Spondylitis
- Ankylosing Spondylitis Disease Activity Score (ASDAS) (out of subjects with presence of psoriatic spondylitis)
- Bath AS Disease Activity Index (BASDAI) (out of subjects with presence of psoriatic spondylitis)
- Morning stiffness (mean of BASDAI Questions 5 and 6)
- Morning stiffness severity 0-10 (BASDAI Question 5)
- Morning stiffness duration 0-10 (BASDAI Question 6)



#### **Patient Report Outcomes at Baseline**

- Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue
- 36-Item Short Form Health Survey (SF-36) Version 2: physical component summary, mental component summary, and the 8 sub-domain scores
- EuroQol-5D-5L (EQ-5D-5L) index and VAS score
- Work Productivity and Activity Impairment (WPAI)
- Self-Assessment of Psoriasis Symptoms (SAPS)

## Tobacco/Nicotine and Alcohol Use

- Tobacco/Nicotine Use [user, ex-user, non-user, unknown]
- Alcohol Use [drinker, ex-drinker, non-drinker, unknown]

## 6.2 Medical History

Medical history data will be summarized and presented for FAS population using body systems and conditions/diagnoses as captured on the CRF. The body systems will be presented in alphabetical order and the conditions/diagnoses will be presented in alphabetical order within each body system. The number and percentage of subjects with a particular condition/diagnosis will be summarized for each randomized treatment group as well as overall. Subjects reporting more than one condition/diagnosis within a body system will be counted only once for that body system. No statistical comparison will be performed for medical history reporting.

#### 6.3 Prior Treatment and Concomitant Medications

Prior and concomitant medications will be summarized by each randomized treatment group as well as overall for FAS. Prior medications are those medications taken prior to the first dose of study drug. This includes medications with a start date before the first study drug administration date, regardless of the end date of these medications. Medications taken on the day of the first dose of study drug are not counted as prior medications. Concomitant medications are those medications, other than study drug,



taken after the first dose of study drug and within 1 day of the last dose of study drug. This includes medications with a start date between first study drug administration and last study drug administration + 1 day, as well as, medications with a start date prior to first dose of study drug and which are ongoing after first dose of study drug. Medications taken on the day of the first dose of study drug are counted as concomitant medications.

The number and percentage of subjects who received a prior medication and the number and percentage of subjects who received a concomitant medication will be tabulated separately by the generic name assigned by the most current version of the World Health Organization (WHO) Drug Dictionary.

#### 6.4 Protocol Deviations

Protocol deviations based on ICH deviation criteria are categorized as follows:

- 1. Those who entered the study even though they did not satisfy the entry criteria
- 2. Those who developed withdrawal criteria during the study and were not withdrawn
- 3. Those who received the wrong treatment or incorrect dose, and
- 4. Those who received an excluded or prohibited concomitant medication.

The protocol deviations listed above will be summarized and listed by treatment group.

## 7.0 Patient Disposition

The following will be summarized by randomized treatment group as well as overall:

- number of subjects randomized,
- number of subjects included in key analysis populations (Full Analysis Set and Per Protocol Analysis Set for efficacy analysis, Safety Analysis Set for safety analysis),
- number of subjects who completed Period 1 study participation,
- number of subjects who entered Period 2,

• number of subjects who completed overall study (Period 1 and Period 2) participation (if applicable).

Premature discontinuation details will be further summarized separately for Period 1 and Period 2 as follows.

#### Period 1

The number and percentage of subjects who completed Period 1 and prematurely discontinued in Period 1 will be summarized by randomized treatment group, separately by study drug completion/discontinuation and by study participation completion/discontinuation, with the reason for discontinuation collected from the CRF by the following categories:

- Adverse event (AE)
- Withdrew consent
- Lost to follow-up
- Lack of efficacy
- Other.

In addition, the number and percentage of subjects entered Period 2 will be summarized by randomized treatment group.

For Week 24 reporting, this summary will also be presented for study drug completion/discontinuation by Week 24.

### Period 2

Period 2 patient dispositions and reason for discontinuation will be summarized with the same categories as given above for Period 1 for overall total and by treatment in Period 2, defined as follows:

1. Upadacitinib 15 mg QD



#### 2. Upadacitinib 30 mg QD

Among the subjects who entered Period 2 participation (regardless of whether subject entered Period 2 on study drug), the number and percentage of subjects who completed and prematurely discontinued study participation in Period 2 will be summarized.

Among the subjects who entered Period 2 on study drug, the number and percentage of subjects who completed and prematurely discontinued study drug in Period 2 will be summarized.

### Summary of Dose Switch from Upadacitinib 30 mg QD to 15 mg QD

Starting with Amendment 7.01.01 (for Japan) and Amendment 8 and 8.01 (for global), subjects receiving upadacitinib 30 mg QD will be switched to upadacitinib 15 mg QD. The visit at which dose switch occurs could be different for each subject. For subjects on upadacitinib 30 mg QD in Period 2, the number and percentage of subjects switching to upadacitinib 15 mg QD at each visit will be summarized.

## 8.0 Study Drug Exposure and Compliance

## 8.1 Study Drug Exposure

For short term up to Week 24, the duration of exposure to study drug will be summarized for the safety analysis set by the randomized treatment groups.

For long term, the duration of exposure to study drug will be summarized for the safety analysis set by the following groups.

## 1. Upadacitinib 15 mg QD

This includes upadacitinib 15 mg QD exposure from subjects starting on upadacitinib 15 mg QD and subjects switching from placebo to upadacitinib 15 mg QD.

#### 2. Upadacitinib 30 mg QD



This includes upadacitinib 30 mg QD exposure from subjects starting on upadacitinib 30 mg QD and subjects switching from placebo to upadacitinib 30 mg QD. Exposure is censored at time of dose switch from upadacitinib 30 mg QD to upadacitinib 15 mg QD.

Upadacitinib 15 mg QD switched from upadacitinib 30mg QD
 This includes upadacitinib 15 mg QD exposure from subjects who switched dose from upadacitinib 30 mg QD to upadacitinib 15 mg QD.

Starting with Amendment 7.01.01 (for Japan) and Amendment 8 and 8.01 (for global), subjects receiving upadacitinib 30 mg QD will be switched to receiving upadacitinib 15 mg QD. Exposure to upadacitinib 30 mg QD (Groups 2) will be censored prior to the day subject received the first dose of upadacitinib 15 mg QD, and subsequent exposure to upadacitinib 15 mg QD will be summarized under a separate group (Group 3).

Exposure to upadacitinib and placebo is defined as last dose date minus first dose date plus 1 day.

The duration of exposure to study drug will be summarized for each group as specified above, with the number of subjects, mean, standard deviation, median, minimum and maximum values. In addition, the number and percentage of subjects exposed to study drug will be summarized for the following cumulative duration intervals.

- $\geq 2$  weeks
- $\geq 1$  month
- $\geq 3$  months
- $\geq$  6 months
- > 9 months
- $\geq 12$  months
- $\geq 18$  months
- $\geq 2$  years

- $\geq 2.5$  years
- $\geq 3$  years
- $\geq 3.5$  years
- $\geq$  4 years
- $\geq 4.5$  years
- $\geq$  5 years
- $\geq 5.5$  years

## 8.2 Compliance

Study drug compliance will be summarized for each treatment group at Week 24. The compliance is defined as the number of tablets taken (i.e., the difference between the number of tablets dispensed and the number of tablets returned) during the subject's participation up to Week 24 divided by the number of days that the subject was in the Treatment Phase up to Week 24.

## 9.0 Efficacy Analysis

#### 9.1 General Considerations

There are two sets of planned efficacy analysis: efficacy analysis through Week 24 and long-term efficacy analysis. Unless otherwise noted, all efficacy analyses will be carried out using the FAS population.

## 9.1.1 Efficacy Analysis at Different Phases of the Study

#### Efficacy Analysis Through Week 24

Efficacy analysis by randomized treatment groups (upadacitinib 15 mg QD, upadacitinib 30 mg QD and the combined placebo group) will be performed on efficacy data up to Week 24. No protocol-defined treatment switching will occur prior to the time point. Formal statistical inference will be generated, and results from this set of analysis will be used as the key efficacy findings of this study.



#### **Long-Term Efficacy Analysis**

Long-term efficacy analysis will be performed on As Observed data (defined in Section 9.1.2) by randomized treatment group sequence as described below:

- 1. Placebo → Upadacitinib 15 mg QD
- 2. Placebo → Upadacitinib 30 mg QD
- 3. Upadacitinib 15 mg QD
- 4. Upadacitinib 30 mg QD

Descriptive statistics and 95% confidence intervals will be provided for all treatment sequences.

For long term efficacy analysis, subjects will continue to be summarized under the treatment sequences as described above, regardless of dose switch from upadacitinib 30 mg QD to upadacitinib 15 mg QD – i.e., for treatment sequences 2 and 4, data collected after dose switch will continue to be summarized under the same treatment sequences. The visit at which dose switch occurs could be different for each subject. The first and last visits at which dose switch occurs will be noted in the summary. In addition, sensitivity analyses will be performed where the subjects who switched from upadacitinib 30 mg QD to 15 mg QD will be censored at the time of dose switch, and efficacy values before & post switch will be summarized separately.

## 9.1.2 Handling of Missing Data and Intercurrent Events

#### Non-Responder Imputation (NRI) Approach

The NRI approach will handle data for binary endpoints as follows.

• Subjects who prematurely discontinue from study drug will be considered as non-responders for all subsequent visits after discontinuation.



• In addition, any subject with any missing value for the binary endpoints at a specific visit will be treated as non-responder for that visit.

NRI data handling will be used for the primary estimand (refer to Section 9.2.1) for the binary endpoints.

#### Mixed-Effects Model Repeated Measures (MMRM) Up to Week 24

The repeated measure analysis will be conducted using mixed models including observed data at all visits. For the MMRM analysis, data collected after premature discontinuation of study drug will be excluded. The mixed model includes the categorical fixed effects of treatment, visit, treatment-by-visit interaction, the stratification factor current DMARD use (yes/no) and the continuous fixed covariates of baseline measurement. An unstructured variance covariance matrix will be used. The parameter estimations are based on the assumption of data being missing at random (MAR) and using the method of restrictive maximum likelihood (REML). MMRM will be used for the primary estimand of key continuous endpoints (refer to Section 9.2.3).

#### As Observed (AO)

The AO data handling will not impute values for missing evaluations, and thus a subject who does not have an evaluation on a scheduled visit will be excluded from the AO analysis for that visit. Regardless of premature discontinuation of study drug or use of rescue medication, all observed data will be used in the analysis. The AO data handling will be used to facilitate the supplementary analysis for both binary and continuous endpoints (refer to Section 9.2.2 and Section 9.2.3 where the corresponding supplementary estimands for the primary and ranked secondary endpoints are described respectively).

The intent-to-treat (ITT) principle for the analysis using AO data, AO (with imputation), where additional missing data will be imputed as non-responders, will be used for the



supplementary analysis of the primary and key secondary binary endpoints. AO with imputation will not be provided for Week 104 analysis and future analyses.

## <u>Mixed Effect Model Repeat Measurement (MMRM) and Generalized Linear Mixed Model (GLMM) for Long-Term Analysis</u>

The repeated measure analysis will be conducted using mixed model including As Observed measurements at all visits. MMRM will be used for continuous endpoints and GLMM will be used for binary endpoints. The mixed models will include the categorical fixed effects of treatment, visit and treatment-by-visit interaction, and stratification factor current DMARD use (yes/no). The categorical fixed effect of subject's discontinuation status may also be included in the model as appropriate. For the MMRM analysis of change from baseline in continuous endpoints, the baseline measurement will be included as a continuous fixed covariate. Unstructured, Toeplitz, compound symmetry, or other covariance structures may be considered.

## 9.2 Efficacy Analysis Through Week 24

## 9.2.1 Primary Efficacy Analysis of the Primary Efficacy Endpoint

The primary efficacy endpoint is ACR20 response at Week 12. The primary estimand is the difference in the proportion of PsA patients who achieved ACR20 response at Week 12 and did not discontinue study drug by Week 12, comparing those who are randomized to each upadacitinib dose group and received study drug to those who are randomized to placebo and received study drug.

Analysis of the primary endpoint will be conducted on the FAS based on randomized treatment groups (upadacitinib 15 mg QD, upadacitinib 30 mg QD versus the combined placebo groups). Point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Comparisons of the primary endpoint will be made between each upadacitinib dose and the combined placebo group using the Cochran-Mantel-Haenszel test (CMH) (refer to Appendix A) adjusting for the main stratification factor of current DMARD use (yes/no). Point estimate, 95% CI



using normal approximation and p-value for the treatment comparison will be presented. Nominal p-values constructed using the CMH test will be provided. The multiplicity adjusted (as described in Section 9.2.5) testing results will also be provided. NRI data handling will be used to facilitate the primary estimand. In addition, the number and percentage of non-responders by the intercurrent events, such as discontinuation of study drug prior to or at Week 12 or missing Week 12 ACR measurement will be summarized.

## 9.2.2 Supplementary Analysis of the Primary Efficacy Endpoint

For the primary efficacy endpoint, the same CMH analysis as detailed in Section 9.2.1 will be repeated using As Observed (AO) data handling without any imputation as supplementary analysis. This will be conducted on the FAS based on randomized treatment groups. The corresponding estimand for the supplementary analysis is the difference in the proportion of PsA patients who achieved ACR20 response at Week 12, regardless of whether the subject had discontinued study drug by Week 12, comparing each upadacitinib dose group vs placebo. The analysis will be conducted for those who are randomized, received study drug and have the efficacy measurement at Week 12 visit.

In addition to the supplementary analysis based on AO data, to explore various missing data assumptions including missing not at random (MNAR), tipping point analysis will also be performed for the primary endpoint by multiple imputations using logistic regression, allowing the imputed ACR response rate to systematically vary from 0% to 100% in both upadacitinib and placebo, respectively. Details of the tipping point analysis are outlined in Appendix B. Supportive analysis will also be conducted on the Per Protocol Analysis Set using the CMH model and NRI data handling.

## 9.2.3 Key Secondary Efficacy Analyses

The following is a list of ranked key secondary endpoints:

1. Change from baseline in HAQ-DI at Week 12;



- Static Investigator Global Assessment (sIGA) of Psoriasis of 0 or 1 and at least a 2-point improvement from baseline at Week 16 (for subjects with baseline sIGA ≥ 2);
- 3. Psoriasis Area Severity Index (PASI) 75 response at Week 16 (for subjects with ≥ 3% BSA psoriasis at baseline);
- 4. Change from baseline in SF-36 PCS at Week 12;
- 5. Change from baseline in FACIT-Fatigue at Week 12;
- 6. Proportion of subjects achieving Minimal Disease Activity (MDA) at Week 24;
- 7. Change from baseline in Self-Assessment of Psoriasis Symptoms (SAPS) at Week 16.

Additional key secondary efficacy endpoints are:

- 1. ACR50/70 response at Week 12;
- 2. ACR20 response at Week 2.

#### Binary Endpoints

For binary endpoints, frequencies and percentages will be reported for each treatment group. For the ranked secondary endpoints at the time point of interest, the primary estimand is the same as that for the primary efficacy endpoint as defined in Section 9.2.1, except for the definition of the efficacy measurement.

For secondary endpoints applicable only for sub-populations, the estimands will be constructed similarly but based on the subject sub-population, as defined in the below table.



| Endpoint | Sub-population |
|---|---|
| Static Investigator Global Assessment (sIGA) of Psoriasis of 0 or 1 and at least a 2-point improvement from baseline at Week 16 | Subjects with baseline sIGA $\geq 2$ are included in the analysis |
| Psoriasis Area Severity Index (PASI) 75 response at Week 16 | Subjects with $\geq$ 3% BSA psoriasis at baseline are included in the analysis |

For MDA at Week 24, in addition to the NRI data handling as defined in Section 9.1.2, subjects who meet the rescue criteria (i.e., not achieving at least 20% improvement in either or both tender joint count (TJC) and swollen joint count (SJC) at both Week 12 and Week 16) will also be treated as non-responders. The corresponding primary estimand is the difference in the proportion of patients who achieved MDA at Week 24, and who did not discontinue study drug and did not initiate rescue therapy by Week 24. The comparison is for each upadacitinib dose group vs placebo for patients randomized and treated with at least one dose of study drug. Supplementary analysis using AO data handling will also be conducted for binary endpoints. The corresponding supplementary estimand is the same as defined in Section 9.2.2 except for the definition of the efficacy measurement.

Point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Treatment comparisons will be made between each upadacitinib dose and the combined placebo group using the Cochran-Mantel-Haenszel test (refer to Appendix A). The CMH test adjusts for the main stratification factor of current DMARD use (yes/no). Point estimate, 95% CI using normal approximation and the p-value for the treatment difference will be presented.

#### **Continuous Endpoints**

For continuous endpoints, the estimand is the difference in mean change from baseline at the protocol defined time point (e.g., HAQ-DI at Week 12) under the assumption that patients with missing data, including those due to premature discontinuation of study drug, can have their measurements at the protocol defined time point predicted by their



observed data and the observed data for other patients for their respective assessments during follow-up. The comparison is for each upadacitinib dose group vs placebo for patients randomized and treated with at least one dose of study drug.

To analyze the primary estimand for the continuous ranked secondary efficacy endpoints, statistical inference will be conducted using the MMRM model and the associated data handling as described in Section 9.1.2, with fixed effects of treatment, visit, treatment-by-visit interaction, the stratification factor of current DMARD use (yes/no) and the continuous fixed covariate of baseline measurement. The LS mean and 95% CI for each randomized treatment group and the LS mean treatment difference, the associated 95% CI and the p-value between each upadacitinib dose group and the combined placebo group will be provided.

The supplementary analysis for ranked secondary continuous endpoints will be conducted using AO data handling and using the analysis of covariance (ANCOVA) model with treatment and the stratification factor of current DMARD use (yes/no) as the fixed factors and the corresponding baseline values as the covariates. The corresponding estimand is the difference in the mean change from baseline in the efficacy endpoints at the protocol defined time point regardless of treatment discontinuation or use of rescue medication, comparing each upadacitinib dose group vs placebo. The analysis will be conducted for those who are randomized, received study drug and have the efficacy measurement at the protocol defined time point.

For the key continuous endpoint change from baseline in HAQ-DI at Week 12, tipping point analysis will also be conducted using multiple imputation (MI) as additional supplementary analysis to explore various missing data assumptions including missing not at random (MNAR). Details of the tipping point analysis for continuous endpoints are outlined in Appendix C.



## 9.2.4 Efficacy Analyses for Additional Endpoints

Additional efficacy analysis includes the following endpoints at the scheduled time points other than those specified for the primary and key secondary variables:

- Change from baseline in individual components of ACR response
- Change from baseline in Tender Joint Count (TJC) (0-68);
- Change from baseline in Swollen Joint Count (SJC) (0-66);
- Change from baseline in Physician Global Assessment (PGA) Disease Activity (NRS);
- Change from baseline in Patient's Global Assessment (PtGA) Disease Activity (NRS);
- Change from baseline in Patient's Assessment of Pain Numerical Rating Scale (NRS);
- Change from baseline in Health Assessment Questionnaire Disability Index (HAQ-DI);
- Change from baseline in High-Sensitivity C Reactive Protein (hs-CRP);
- ACR 20/50/70 response rates;
- Proportion of subjects achieving MDA;
- Change from baseline in Leeds Dactylitis Index (LDI) (for subjects with baseline LDI > 0);
- Change from baseline in dactylitis count (for subjects with baseline LDI > 0);
- Proportion of subjects with resolution of dactylitis (defined as LDI = 0) (for subjects with baseline LDI > 0);
- Change from baseline in LEI (for subjects with baseline LEI > 0);
- Proportion of subjects with resolution of enthesitis defined as LEI = 0 (for subjects with baseline LEI > 0);
- Change from baseline in SPARCC Enthesitis Index (for subjects with baseline SPARCC Enthesitis Index > 0);
- Proportion of subjects with resolution of enthesitis defined as SPARCC
   Enthesitis Index = 0 (for subjects with baseline SPARCC Enthesitis Index > 0);



- Change from baseline in total enthesitis count (for subjects with baseline total enthesitis count > 0);
- Proportion of subjects with resolution of enthesitis defined as total enthesitis count = 0 (for subjects with baseline total enthesitis count > 0);
- PASI 75/90/100 response rates (for subjects with ≥ 3% Body Surface Area (BSA) psoriasis at baseline);
- Proportion of subjects achieving a static Investigator Global Assessment of psoriasis (sIGA) score of 0 or 1 and at least a 2-point improvement from baseline (for subjects with baseline sIGA ≥ 2);
- Change from baseline in BSA-Ps (for subjects with baseline BSA > 0%);
- Modified Psoriatic Arthritis Response Criteria (PsARC) response rate;
- Change from baseline in Disease Activity Score 28 (DAS28) (CRP);
- Change from baseline in DAS28 (ESR);
- Change from baseline in PsA Disease Activity Score (PASDAS);
- Change from baseline in Disease Activity In Psoriatic Arthritis (DAPSA) score;
- Change from baseline in Short Form 36 (SF-36) Health;
- Change from baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue;
- Change from baseline in EuroQol-5D-5L (EQ-5D-5L) index and VAS score;
- Change from baseline in Work Productivity and Activity Impairment (WPAI);
- Cumulative Health Resource Utilization (HRU);
- Change from baseline in Self-Assessment of Psoriasis Symptoms (SAPS);
- Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) (out of subjects with presence of psoriatic spondylitis at baseline);
- BASDAI 50 response rates (out of subjects with presence of psoriatic spondylitis at baseline);
- Change from baseline in Morning stiffness (mean of BASDAI Questions 5 and 6)
- Change from baseline in Morning stiffness severity 0 10 (BASDAI Question 5)



- Change from baseline in Morning stiffness duration 0 10 (BASDAI Question 6)
- Change from baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) (out of subjects with presence of psoriatic spondylitis at baseline);
- Proportion of subjects with ASDAS Inactive Disease (out of subjects with presence of psoriatic spondylitis at baseline);
- Proportion of subjects with ASDAS Major Improvement (out of subjects with presence of psoriatic spondylitis at baseline);
- Proportion of subjects with ASDAS Clinically Important Improvement (out of subjects with presence of psoriatic spondylitis at baseline);
- Proportion of subjects achieving a clinically meaningful improvement in HAQ-DI (≥ 0.35).

For binary endpoints, frequencies and percentages will be reported for each treatment group. NRI will be used for primary analysis. AO will be used as supplementary analysis. Point estimate and 95% CI using normal approximation will be provided for the response rate for each randomized treatment group. Treatment comparisons will be made between each upadacitinib dose to the combined placebo group using the CMH (refer to Appendix A) test adjusting for the main stratification factor of current DMARD use (yes/no). Point estimate, 95% CI using normal approximation and the nominal p-value for the treatment difference will be presented.

For continuous endpoints, the LS mean and 95% CI for each randomized treatment group and the LS mean treatment difference, the associated 95% CI and the p-value between each upadacitinib dose group and the combined placebo group will be provided using MMRM model as described in Section 9.2.3, with fixed effects of treatment, visit, treatment-by-visit interaction, the stratification factor of current DMARD use (yes/no) and the continuous fixed covariates of baseline measurement. The nominal p-value will be provided.

For change from baseline in each of the seven ACR components, the ANCOVA model using AO data handling as described in Section 9.2.3 will be conducted as supplementary



analysis, with treatment and the stratification factor of current DMARD use (yes/no) as the fixed factors and the corresponding baseline values as the covariates. Nominal p-values will be provided.

## 9.2.5 Handling of Multiplicity

The overall type I error rate of the primary and ranked key secondary endpoints for the two doses will be strongly controlled using a graphical multiple testing procedure. Specifically, the testing will utilize the endpoint sequence of primary endpoint followed by the ranked key secondary endpoints in the order as specified in Section 9.2.3, and will begin with testing the primary endpoint using  $\alpha$  of 0.025 for each dose. Continued testing will follow a pre-specified  $\alpha$  transfer path which includes downstream transfer along the endpoint sequence within each dose as well as cross-dose transfer. Adjusted p-values for the primary and ranked key secondary endpoints will be provided based on the testing procedure.

The graph for the testing procedures is provided in Figure 2. In the graph, the arrows specify the α transfer paths. Once an endpoint is rejected (i.e., deemed significant) at its assigned significance level, its significance level will be transferred to subsequent endpoint(s) following the arrow(s). The numbers on the arrows denote the weights for transferring significance levels. Specifically, the weight 1 denotes 100% transfer of significance level.

Figure 2. Graphical Multiple Testing Procedure




#### 9.2.6 Efficacy Subgroup Analysis

The primary efficacy endpoint will be examined in the subgroups listed in Table 6 below. Treatment difference between each upadacitinib dose and the combined placebo group will be presented with point estimate and 95% confidence interval using normal approximation. No p-value will be provided for subgroup analysis.

**Table 6.** Subgroups for Efficacy Analysis

| Subgroup Factor | Categories |
|---|---|
| Age | $<65, \ge 65 - <75, \ge 75$ years (if sample size allows) |
| Sex | Male or Female |
| BMI | $< 25 \text{ kg/m}^2 \text{ or} \ge 25 \text{ kg/m}^2$ |
| Race | White, Non-white |
| Geographic region | North America, Western Europe and Oceania, Eastern<br>Europe, Latin-America, Asia, and Other |
| Duration of PsA diagnosis | $\leq 5, > 5 - \leq 10 > 10$ years |
| Baseline hsCRP | $\leq$ ULN or $>$ ULN |
| Number of prior failed biologic DMARDs | = 1, > 1 |
| Current use of non-biologic DMARDs | Yes or No |

### 9.3 Long-Term Efficacy Analysis

Assessments to evaluate long-term efficacy will be analyzed for the following measures at Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 44, 56 and every 12 weeks thereafter until completion of the study:

- ACR20/50/70 response rates
- Change from baseline in individual ACR components
- Change from baseline in DAS28 (CRP) and DAS28 (ESR)
- PsARC response rate
- Change from baseline in DAPSA
- Proportion of subjects achieving a clinically meaningful improvement in HAQ-DI (≥ 0.35)



Assessments to evaluate long-term efficacy will be analyzed for the following measures at Week 12, 24, 36, 56 and every 12 weeks thereafter until completion of the study:

- Change from baseline in EQ-5D-5L index and VAS score
- Change from baseline in FACIT-Fatigue
- Change from baseline in SF-36
- Change from baseline in WPAI
- Change from baseline in BASDAI
- Cumulative HRU
- Change from baseline in PASDAS
- BASDAI 50 response rates
- Change from baseline in ASDAS
- Proportion of subjects with ASDAS Inactive Disease
- Proportion of subjects with ASDAS Major Improvement
- Proportion of subjects with ASDAS Clinically Important Improvement

Assessments to evaluate long-term efficacy will be analyzed for the following measures at Week 12, 16, 24, 36, 56 and every 12 weeks thereafter until completion of the study:

- Change from baseline in BSA-Ps
- PASI 75/90/100 response rates
- Static Investigator Global Assessment (sIGA) of Psoriasis of 0 or 1 and at least a 2-point improvement from baseline
- Proportion of subjects achieving Minimal Disease Activity (MDA)
- Change from baseline in LDI
- Change from baseline in LEI
- Change from baseline in SPARCC enthesitis index
- Change from baseline in dactylitis count
- Proportion of subjects with resolution of dactylitis
- Proportion of subjects with resolution of enthesitis sites included in the LEI



- Proportion of subjects with resolution of enthesitis sites included in the SPARCC Enthesitis Index
- Change from baseline in total enthesitis count
- Proportion of subjects with resolution of enthesitis

Assessments to evaluate long-term efficacy will be analyzed for the following measures at Week 16, 24, 36, 56 and every 12 weeks thereafter until completion of the study:

• Change from baseline in SAPS

Descriptive statistics based on AO data will be provided for each randomized treatment group sequence as defined in Section 9.1.1. These include the number of observations, mean, standard deviation, 95% CI, median, minimum, and maximum for continuous endpoints; and frequencies and percentages with 95% CI using normal approximation for binary endpoints.

In addition, NRI approach and/or GLMM will be used for binary endpoint analysis, and MMRM will be used for continuous endpoint analysis. The analyses will be performed for the treatment sequences. The longitudinal analysis using MMRM or GLMM was described in Section 9.1.2. Point estimates and 95% CI from the model will be provided for each treatment sequence. Plot for each randomized treatment group sequence over time will be provided for key endpoints.

#### 9.4 Efficacy Variables Definitions and Conventions

#### 9.4.1 ACR Criteria

ACR criteria are a commonly used standard criteria set mentioned in the FDA industry guidance to evaluate the effectiveness of investigational drug in reduction of disease activity. It is a composite measurement calculated based on the improvement over a set of core measurements.



ACR20 is defined as at least 20% improvement (compared to baseline values) in tender and swollen joint counts and at least 20% improvement in 3 of the remaining 5 core set measures (subject assessment of pain, subject global assessment of disease activity, physician global assessment of disease activity, subject assessment of physical function and acute phase reactant hsCRP).

ACR50 and ACR70 are similarly defined with at least 50% and 70% improvement, respectively.

A subject will be classified as an ACR20 (ACR50, ACR70) responder, if the following conditions are met:

- 1.  $\geq$  20% (50%, 70%) improvement from baseline in tender joint count (TJC68) and
- 2.  $\geq$  20% (50%, 70%) improvement from baseline in swollen joint count (SJC66) and
- 3.  $\geq 20\%$  (50%, 70%) improvement from baseline in at least 3 of the following 5:
  - patient's assessment of pain
  - patient's global assessment of disease activity (PtGA)
  - physician's global assessment of disease activity (PGA)
  - patient's self-assessment of physical function (i.e., measured by Health Assessment Questionnaire HAQ-DI score)
  - Acute-phase reactant value high-sensitivity CRP (hsCRP)

Seven components are included in the ACR response criteria. Missing values for a component can occur due to data collection issues for a particular form, a missed visit or dropout from the study. Depending on the pattern of the missing components, ACR responses may be or may not be determined for a visit date using (partially) observed values only. In the case when ACR responses cannot be determined for any visit date within a visit window, partially observed data from different visit dates within the same visit window can be combined to determine ACR responses for the visit window.

To maximize the utilization of observed information at certain visits and be scientifically as robust as possible, the principle to calculate ACR response is to minimize imputation whenever possible. "As Observed" ACR response will be calculated first based on a derived visit window instead of the nominal visit identifier (e.g., Week 6 visit) collected from the CRF.

To calculate "as observed" ACR responses:

Identify the observed component 20% improvement indicator (0/1/missing), 1 means achieving  $\geq$  20% improvement from baseline and 0 means < 20% improvement from baseline.

ACR20 = 0 if TJC indicator = 0 OR SJC indicator = 0 OR at least 3 out of 5 components improvement indicators = 0;

ACR20 = 1 if TJC indicator = 1 AND SJC indicator = 1 AND at least 3 out of 5 components improvement indicators = 1

For all other cases, "as observed" ACR20 = missing since ACR20 cannot be determined.

The following table illustrates examples for observed ACR calculations.

| Example | TJC<br>68 | SJC<br>66 | Component 1 | Component 2 | Component 3 | Component 4 | Component 5 | ACR20-<br>Response? |
|---|---|---|---|---|---|---|---|---|
| A | 1 | 1 | 1 | 1 | 1 | | | Yes |
| В | 1 | 0 | 1 | 1 | 1 | 1 | 1 | No |
| C | | 0 | | | | | | No |
| D | 1 | | 1 | 1 | 1 | 1 | 1 | |
| E | 1 | 1 | 0 | 0 | 0 | 1 | 1 | No |
| F | | | 0 | 0 | 0 | | | No |
| G | 1 | 1 | 1 | 1 | 0 | 0 | | |

Legend: 1 = 20% improved compared to baseline; 0 = 20% improved compared to baseline; "." Missing

Derived visit windowing Rule for ACR Response Calculation:



To identify the component value in a visit window:

ACR component values will first be determined at each date within a visit window.

ACR component values at each date will be combined to determine the "as observed" ACR composite score at each date in each window.

After this calculation, if multiple non-missing ACR composite scores are available within a given visit window, the non-missing ACR composite score closest to the target day will be used. If two composite scores have the same distance from the target day, the later one will be used. The corresponding date will be used as the "as observed" ACR response date in the derived efficacy dataset.

If a non-missing ACR composite score is not available for any day within a given visit window, the windowed component values for that visit will be used to calculate the ACR composite score for that visit window (component value windowing follow the same rules as in steps described above). Date of TJC will be used as the "as observed" ACR date in the derived efficacy dataset.

The following rules are applied for the NRI imputation for the ACR responses.

Non-Responder Imputation (NRI):

- Step 1: all missing components will be imputed using LOCF, and then the ACR composite score can be calculated
- Step 2: if the ACR composite score cannot be determined by step 1, the ACR composite score will be imputed as 0. In addition, subjects who prematurely discontinue from the study drug will be considered as non-responders (ACR = 0) for all subsequent visits after the discontinuation date.



#### 9.4.2 Joint Evaluation

Anatomical joints are evaluated for swelling and tenderness at every study visit. The 34 anatomical joints in Table 7 are assessed in this study for both the left and right side of the body.

Table 7. Anatomical Joints Assessed for Calculation of Tender and Swollen Joint Counts (TJC68 and SJC66)

| Temporomandibular | Sternoclavicular | Acromio-clavicular | Shoulder |
|---|---|---|---|
| Elbow | Wrist | Metacarpophalangeal I | Metacarpophalangeal II |
| Metacarpophalangeal III | Metacarpophalangeal IV | Metacarpophalangeal V | Thumb Interphalangeal |
| Proximal Interphalangeal II | Proximal<br>Interphalangeal III | Proximal<br>Interphalangeal IV | Proximal Interphalangeal V |
| Distal<br>Interphalangeal II | Distal<br>Interphalangeal III | Distal<br>Interphalangeal IV | Distal<br>Interphalangeal V |
| Hip <sup>a</sup> | Knee | Ankle | Tarsus |
| Metatarsophalangeal I | Metatarsophalangeal II | Metatarsophalangeal III | Metatarsophalangeal IV |
| Metatarsophalangeal V | Great Toe/Hallux | Interphalangeal II | Interphalangeal III |
| Interphalangeal IV | Interphalangeal V | | |

a. Hip joints are not assessed for swelling.

At each study visit, a joint evaluator will assess whether a particular joint was "tender or painful" where presence of tenderness is scored as "1" and the absence of tenderness is scored as "0," provided the joint was not replaced ("9") or could not be assessed ("NA") due to other reasons (e.g., post-corticosteroid joint injection). The total tender joint count (TJC68), which is based on 68 joints, will be derived as the sum of all "1s" and proportional extrapolation will be used to impute joint counts for the joints that are replaced or not assessed. A similar method will be followed for the derivation of total swollen joint count (SJC66), which is based on 66 joints as the hip joints are excluded. Thus, the range for TJC68 will be 0 to 68 and 0 to 66 for SJC66.

# 9.4.3 Patient's Global Assessment of Disease Activity Numeric Rating Scale (NRS)

The subject will assess his/her disease activity using the Patient's Global Assessment of Disease NRS. The range is 0 to 10 with no activity being indicated by 0 and severe activity by 10.

# 9.4.4 Physician's Global Assessment of Disease Activity Numeric Rating Scale (NRS)

The physician will assess Patient's disease activity at the time of visit using the Physician's Global Assessment of Disease NRS. The range is 0 to 10 with no activity being indicated by 0 and severe activity by 10.

#### 9.4.5 Patient's Assessment of Pain Numeric Rating Sale (NRS)

The subject will assess his/her pain using the Patient's Global Assessment Pain NRS. The range is 0 to 10 with no activity being indicated by 0 and severe activity by 10.

### 9.4.6 Disease Activity Score (DAS28)

DAS28 (CRP) and DAS28 (ESR) are composite indices to assess disease activity in PsA using hsCRP or ESR measurement, respectively. The DAS28 provides a score between 0 and 10, indicating arthritis disease activity at the time of measurement.

DAS28 (CRP) and DAS28 (ESR) is calculated based on Tender Joint Count, Swollen Joint Count, PtGA of Disease Activity (0-100), and hsCRP (in mg/L) or ESR (mm/hr).

DAS28 (CRP) = 
$$0.56 \times \sqrt{\text{TJC28*}} + 0.28 \times \sqrt{\text{SJC28**}} + 0.36 \times \ln(\text{hsCRP*} + 1) + 0.014 \times \text{PtGA*} + 0.96$$

DAS28 (ESR) = 
$$0.56 \times \sqrt{\text{TJC28*}} + 0.28 \times \sqrt{\text{SJC28**}} + 0.70 \times \ln(\text{ESR}^{\#}) + 0.014 \times \text{PtGA}^{"}$$

where  $\sqrt{ }$  is square root and ln is natural log.

- \* TJC28 refers to the Subject's total Tender Joint Count out of the provided 28 evaluated joints.
- \*\* SJC28 refers to the Subject's total Swollen Joint Count out of the provided 28 evaluated joints.



- & hsCRP refers to the high-sensitivity c-reactive protein lab value. hsCRP unit in the DAS28 (CRP) equation is expressed as mg/L.
- # ESR refers to the Erythrocyte sedimentation rate. ESR unit in the DAS28 (ESR) equation is expressed as mm/hr.
- » PtGA refers to the Patient's Global Assessment of Disease Activity.

Table 8. Anatomical Joints for DAS28 (CRP) Calculation

| Shoulder | Elbow | Wrist | Thumb Interphalangeal |
|---|---|---|---|
| Metacarpophalangeal I | Metacarpophalangeal II | Metacarpophalangeal III | Metacarpophalangeal IV |
| Metacarpophalangeal V | Proximal<br>Interphalangeal II | Proximal Interphalangeal III | Proximal Interphalangeal IV |
| Proximal<br>Interphalangeal V | Knee | | |

As PtGA of Disease Activity is collected with the scale of 0-10 NRS, the variable needs to be multiplied by 10 before being used the DAS28 formula.

To calculate observed DAS28 scores, the observed component value will be calculated first. Then the components will be included in the calculation per the DAS formula selected. If any observed component is missing in a window, then the observed DAS28 score will be missing.

### 9.4.7 Disease Activity in Psoriatic Arthritis (DAPSA) Score

DAPSA is a continuous endpoint that measures the disease activity in psoriatic arthritis. DAPSA consists of five components: Tender Joint Count 68, Swollen Joint Count 66, Patient's Assessment of Pain (0-10 NRS), PtGA of Disease Activity (0-10 NRS), and hsCRP (in mg/dL).

$$DAPSA = SJC66 + TJC68 + Pt pain (0-10 NRS) + PtGA (0-10 NRS) + hsCRP (in mg/dL)$$

To calculate observed DAPSA scores, the observed component value will be calculated first. Then the components will be included in the calculation per the DAPSA formula. If any observed component is missing in a window, then the observed DAPSA score will be missing.

### 9.4.8 PsA Disease Activity Score (PASDAS)

PASDAS is a continuous scale of combined joint, dactylitis and enthesitis assessments, physician and patient global assessments for arthritis, SF36-PCS, and hsCRP measurements.

PASDAS = 
$$(((0.18 \sqrt{(PGA)}) + 0.159 \sqrt{(PtGA)} - 0.253 \sqrt{(SF36-PCS)} + 0.101 \ln (SJC66 + 1) + 0.048 \ln (TJC68 + 1) + 0.23 \ln (Leeds Enthesitis Index + 1) + 0.37 \ln (Tender Dactylitis Count + 1) + 0.102 \ln (hsCRP + 1) + 2) * 1.5,$$

where  $\sqrt{\ }$  is square root and ln is natural log. PtGA is on the scale of 0-100 and PGA is on the scale of 0-100. As PtGA and PGA are collected with the scale of 0-10 NRS, their values need to be multiplied by 10 before being used in the PASDAS formula.

SF36-PCS is the physical component scale in SF36 instrument. The unit for hsCRP is mg/L.

The tender dactylitis count is based on the dactylitis assessment. The count is calculated by summing the digits with a "presence of tenderness" score = 1.

The Leeds Enthesitis Index (LEI) evaluates enthesitis at 6 most commonly involved entheseal sites, as indicated in the table below. The LEI is calculated by taking the sum of the scores from the 6 sites. The LEI ranges from 0 to 6.

| | | To | Tenderness in Left | | | enderness in | n Right |
|---|---|---|---|---|---|---|---|
| | | YES = 1 | NO = 0 | Not Assessed = NA | <b>YES</b> = 1 | NO = 0 | Not Assessed = NA |
| 1 | Lateral epicondyle | | | | | | |
| 2 | Achilles tendon insertion | | | | | | |
| 3 | Medial femoral condyle | | | | | | |



To calculate observed PASDAS scores, the observed component value will be calculated first. Then the components will be included in the calculation per the PASDAS formula. If any observed component is missing in a window, then the observed PASDAS score will be missing.

# 9.4.9 Disability Index of Health Assessment Questionnaire (HAQ-DI)

HAQ-DI is a self-reported patient outcome measurement. It is calculated as the mean of the scores from 8 following categories with a range 0-3: Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. Higher scores reflect greater disability.

The maximum score for all the questions in each category is considered as the score for the category. The HAQ-DI takes into account the subject's use of aids or devices or assistance in the scoring algorithm for a disability category. For each category there is an AIDS OR DEVICES companion variable that is used to record the type of assistance, if any, a subject uses for his/her usual activities. If aids or devices and/or assistance from another person are checked for a category, the score for this category is set to 2 (much difficulty), if the original score is 0 (no difficulty) or 1 (some difficulty). The HAQ-DI is then calculated by summing the adjusted categories scores and dividing by the number of categories answered. The HAQ-DI cannot be calculated if the subject does not have scores for at least 6 categories.

# 9.4.10 Static Investigator Global Assessment of Psoriasis (sIGA)

The sIGA is a 5 point score ranging from 0 to 4, based on the investigator's assessment of the average elevation, erythema, and scaling of all psoriatic lesions. The assessment is considered "static" which refers to the patients disease state at the time of the assessment, without comparison to any of the patient's previous disease states, whether at Baseline or at a previous visit. A lower score indicates less severe psoriasis (0 = clear, 1 = almost clear, 2 = mild, 3 = moderate and 4 = severe).

A binary clinical endpoint based on sIGA is considered in this study. It is the proportion of subjects achieving a sIGA score of 0 or 1 and at least a 2-point improvement from baseline. This endpoint is calculated among the subjects with baseline sIGA score  $\geq 2$ .

### 9.4.11 Psoriasis Area Severity Index (PASI)

Psoriasis Area Severity Index (PASI) has four anatomic sites – head, upper extremities, trunk, and lower extremities – which are assessed for erythema, induration and desquamation using a 5-point scale:

- 0 = no symptoms
- 1 =slight
- 2 = moderate
- 3 = marked
- 4 = very marked

Based on the extent of lesions in a given anatomic site, the area affected is assigned a numerical value:

- 0 = no involvement
- 1 = < 10%
- $\bullet$  2 = 10% 29%
- 3 = 30% 49%
- 4 = 50% 69%
- 5 = 70% 89%
- 6 = 90% 100%

Since the head, upper extremities, trunk and lower extremities correspond to approximately 10, 20, 30 and 40% of body surface area, respectively; the PASI score is calculated using the formula:



$$PASI = 0.1(E_h + I_h + D_h)A_h + 0.2(E_u + I_u + D_u)A_u + 0.3(E_t + I_t + D_t)A_t + 0.4(E_l + I_l + D_t)A_l$$

where *E*, *I*, *D*, and *A* denote erythema, induration, desquamation, and area, respectively, and *h*, *u*, *t*, and *l* denote head, upper extremities, trunk, and lower extremities, respectively. PASI scores range from 0.0 to 72.0 with the highest score representing complete erythroderma of the severest possible degree. Typically scores of 3 or less represent mild disease, scores over 3 and up and including 15 represent moderate disease and scores over 15 are considered to be associated with severe disease.

If an item is missing, PASI is not scored.

PASI 75 (PASI 50, PASI 90, PASI 100) response is achieved if there is at least a 75% (50%, 90%, 100%) reduction in PASI score ( $\geq$  PASI 75/50/90/100 response) at a visit relative to the Baseline PASI score.

PASI is summarized in subjects with  $\geq$  3% BSA (Body Surface Area) psoriasis involvement at baseline.

### 9.4.12 Minimum Disease Activity for PsA

A patient is classified as in MDA when 5 of the following 7 criteria are met:

- TJC68 ≤ 1
- SJC66 < 1
- $PASI \le 1$  or  $BSA-Ps \le 3\%$
- Patient's assessment of pain  $\leq 1.5 (0 10 \text{ NRS})$
- Patient's Global Assessment of disease activity  $\leq 2 (0 10 \text{ NRS})$
- HAQ-DI score  $\leq 0.5$
- Leeds Enthesitis Index  $\leq 1$

MDA response can be determined if at least 5 of the 7 criteria are met (responder), or if at least 3 of the 7 criteria are not met (non-responder). Selection of multiple MDA



responses within one visit window follows the same rules as ACR. Missing values for each component can occur due to data collection issues for a particular form, a missed visit or dropout from the study. Depending on the pattern of the missing components, MDA responses may be or may not be determined for a visit date using (partially) observed values only. In the case when MDA responses cannot be determined for any visit date within a visit window, partially observed data from different visit dates within the visit window can be combined to determine MDA responses for the visit window.

#### 9.4.13 Self-Assessment of Psoriasis Symptoms (SAPS)

The Self-Assessment of Psoriasis Symptoms (SAPS) contains 11 symptom-focused items. Each item is scored from 0 to 10, with 0 being least severe and 10 being most severe. The total score is generated by summing the 11 items. The total score ranges from 0 to 110.

### 9.4.14 Leeds Dactylitis Index (LDI) and Dactylitis Count

The Leeds Dactylitis Index (LDI) is a score based on finger circumference and tenderness, assessed and summed across all dactylitic digits. The presence of dactylitis digit is defined as at least one affected AND tender digit with circumference increase over reference digit  $\geq 10\%$ . For each of 20 digits of a subject, a digit final score needs to be calculated first. For an unaffected digit, the digit final score is set to be 0. For an affected digit, the digit final score is calculated as (A/B-1)\*100\*C if  $A/B \geq 1.1$ , and digit finals score = 0 if A/B < 1.1, where A denotes the circumference of the digit, B the reference circumference, and C the tenderness score. The reference circumference can be either the circumference of the unaffected contralateral digit if available, or from a reference table if otherwise. LDI is the sum of the digit final scores over all 20 digits.

The dactylitis count will be calculated as the number of digits (hands and feet) with presence of dactylitis. The count ranges from 0 to 20.

The proportion of subjects with resolution of dactylitis is defined as the proportion of subjects with LDI = 0.



# 9.4.15 Leeds and SPARCC Enthesitis Indices and Total Enthesitis Count

For the Spondyloarthritis Research Consortium of Canada (SPARCC) enthesitis index 16 sites are evaluated as indicated in rows 1-8 in the table below. Tenderness on examination is recorded as either present (coded as 1), absent (coded as 0), or not assessed for each site. The SPARCC enthesitis index is calculated by taking the sum of the scores from the 16 sites. The SPARCC score ranges from 0 to 16.

The Leeds Enthesitis Index evaluates enthesitis at the 6 entheseal sites indicated in rows 2, 7 and 9 in the table below. Tenderness on examination is recorded as either present (coded as 1), absent (coded as 0), or not assessed for each of the 6 sites. The LEI is calculated by taking the sum of the scores from the 6 sites. The LEI ranges from 0 to 6.

The total enthesitis count is calculated by taking the sum of the tenderness scores from all 18 sites in the table below.

The proportion of subjects with resolution of enthesitis sites included in the LEI is defined as the proportion of subjects with LEI = 0; the proportion with resolution of the SPARCC Enthesitis Index and of the total enthesitis count are similarly defined.

| | | Tenderness in Left | | Te | enderness | in Right | |
|---|---|---|---|---|---|---|---|
| | | Present = 1 | Absent = 0 | Not Assessed = NA | Present = 1 | Absent = 0 | Not Assessed = NA |
| 1 | Medial epicondyle | | | | | | |
| 2 | Lateral epicondyle | | | | | | |
| 3 | Supraspinatus insertion into the greater tuberosity of humerus | | | | | | |
| 4 | Greater trochanter | | | | | | |
| 5 | Quadriceps<br>insertion into<br>superior border of<br>patella | | | | | | |
| 6 | Patellar ligament<br>insertion into<br>inferior pole of<br>patella or tibial<br>tubercle | | | | | | |
| 7 | Achilles tendon insertion into calcaneum | | | | | | |
| 8 | Plantar fascia<br>insertion into<br>calcaneum | | | | | | |
| 9 | Medial femoral condyle | | | | | | |

# 9.4.16 Body Surface Area (BSA) – Psoriasis

The subject's right or left hand should be selected as the measuring device. For purposes of clinical estimation, the total surface of the palm plus five digits will be assumed to be approximately equivalent to 1%. Measurement of the total area of involvement by the physician is aided by imagining if scattered plaques were moved so that they were next to each other and then estimating the total area involved.

# 9.4.17 Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and Morning Stiffness Score

The BASDAI is composed of 6 items investigating 5 domains (fatigue, spinal pain, joint pain/swelling, areas of localized tenderness, morning stiffness), with 1 item for each of the first four domains and 2 items for the last domain (morning stiffness). Each item is scored on a 0-10 NRS. A lower score indicates less disease activity.

Scoring of the BASDAI is as follows:

- 1. Measure each item of the BASDAI in NRS (out of a total of 10)
- 2. BASDAI Score = 0.2\*(Item1 + Item2 + Item3 + Item4 + 0.5\*Item5 + 0.5\*Item6)

The BASDAI Score ranges from 0-10. If one of the 5 items (Questions 1-Question 4, inflammation) is missing, then the score is the mean of the 4 non-missing items (total of 4 non-missing items divided by 4). If more than 1 of the 5 items is missing, then the BASDAI score is missing.

Note: Question 5 and Question 6 jointly constitute Item 5 (inflammation). If both Questions 5 and 6 are missing, and questions 1 through 4 are non-missing, then only one item will be considered missing. The BASDAI score can still be calculated as the mean of Questions 1 – 4. However, if, for example, both Question 6 and Question 1 are missing, then 2 items will be considered missing, as the inflammation calculation would be incomplete. The BASDAI score would then be considered missing in this case.

The Morning Stiffness Score is the average of BASDAI questions 5 and 6 and it ranges from 0-10.

#### 9.4.18 Modified Psoriatic Arthritis Response Criteria (PsARC)

The modified PsARC is a PsA-specific composite responder index. To achieve response, a subject must achieve 2 of the following 4 items, one of which has to be a Tender Joint Count 68 or Swollen Joint Count 66, and no worsening of any measure:

- $\geq 30\%$  improvement in TJC68
- $\geq 30\%$  improvement in SJC66
- Improvement in PtGA of Disease Activity NRS
- Improvement in PGA of Disease Activity NRS

Four components are included in the PsARC criteria. Missing values for each component can occur due to data collection issues for a particular form, a missed visit or dropout from the study. In the case when PsARC responses cannot be determined for any visit date within a visit window, partially observed data from different visit dates within the visit window can be combined to determine PsARC responses for the visit window.

#### 9.4.19 Ankylosing Spondylitis Disease Activity Score (ASDAS)

Parameters used for the calculation of ASDAS:

- 1. Patient's assessment of total back pain (BASDAI Question 2)
- 2. PtGA of disease activity (0-10 NRS)
- 3. Peripheral pain/swelling (BASDAI Question 3)
- 4. Duration of morning stiffness (BASDAI Question 6)
- 5. High-sensitivity C-reactive protein (hs-CRP) in mg/L.

#### Calculation of ASDAS:

$$ASDAS_{hs\text{-}CRP} = 0.121 \times total \ back \ pain + 0.110 \times PtGA + 0.073 \times peripheral \\ pain/swelling + 0.058 \times duration \ of \ morning \ stiffness + 0.579 \times \\ Ln(hs\text{-}CRP+1).$$

To calculate observed ASDAS scores, the observed component value will be calculated first. Then the components will be included in the calculation per the ASDAS formula. If any observed component is missing in a window, then the observed ASDAS score will be missing.



ASDAS score is categorized by the following ASDAS Disease Activity States:

• ASDAS Inactive Disease: ASDAS < 1.3

• ASDAS Moderate Disease:  $1.3 \le ASDAS < 2.1$ 

• ASDAS High Disease:  $2.1 \le ASDAS \le 3.5$ 

• ASDAS Very High Disease: ASDAS > 3.5

ASDAS Response categories are defined as follows:

- ASDAS Major Improvement (a change from baseline  $\leq$  -2.000)
- ASDAS Clinically Important Improvement (a change from baseline  $\leq -1.100$ )

#### 9.4.20 FACIT-Fatigue Questionnaire (FACIT-F)

The FACIT Fatigue Questionnaire is a 13-item tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point scale (4 = not at all fatigued to 0 = very much fatigued). The Fatigue scale ranges from 0 to 52, with higher scores indicating less fatigue.

Item score for each item is calculated by either subtracting from 4 or adding 0 depending on whether it is a reversal item or not. FACIT Fatigue Scale is then calculated by adding up all item scores, multiplying by 13 and dividing by the number of items answered. If less than 7 items are answered, the scale will not be computed.

#### 9.4.21 EuroQoL-5D (EQ-5D-5L)

EQ-5D measures 5 dimensions of health status (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) with 5 levels per dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems corresponding to Level 1 to Level 5 respectively) and includes the EQ Visual Analogue Scale (EQ VAS). The 5 dimensions of health status are converted into a single index value. The change from baseline of the index value and the EQ VAS will be analyzed and reported. UK scoring algorithm will be used.



#### 9.4.22 Form SF-36v2

The 36-Item Short Form, Version 2 (SF-36v2) health survey consists of 36 general health questions. It has 2 components: physical and mental. For each component, a transformed summary score is calculated using 8 sub domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.

The coding and scoring for the SF-36 will use the software provided by QualityMetrics.

# 9.4.23 Work Productivity and Activity Impairment Questionnaire Psoriatic Arthritis (WPAI)

The Work Productivity and Activity Impairment Questionnaire: Psoriatic Arthritis, V2.0 (WPAI) was developed to measure the effect of overall health and specific symptoms on productivity at work and outside of work. It consists of 6 questions. A lower WPAI score indicates an improvement. The WPAI is collected at the designated study visits listed in the protocol. The WPAI coding and scoring methods are described in the following:

The 6 measures will be derived based on the responses from the 6 questions. The 4 main impairment scores (S1 to S4) are expressed as *percent impairment* based on the 6 questions.

#### **Scores:**

- S0. Employment: defined below in missing data handling conventions
- S1. Absenteeism: Percent work time missed due to PsA:

$$100 \times \left[ \frac{Q2}{Q2 + Q4} \right]$$



S2. Presenteeism: Percent impairment while working due to PsA:

$$100 \times \left\lceil \frac{Q5}{10} \right\rceil$$

S3. Percent overall work impairment due to PsA:

$$100 \times \left[ \frac{Q2}{Q2 + Q4} + \left\{ 1 - \frac{Q2}{Q2 + Q4} \right\} \times \frac{Q5}{10} \right]$$

S4. Percent activity impairment due to PsA:

$$100 \times \left\lceil \frac{Q6}{10} \right\rceil$$

S5. Did subject miss work (defined below). This is needed to derive the proportion of subjects who missed work.

#### **Missing Data Handling Conventions**

When calculating the WPAI: PsA scores, the following computational notes should be followed.

- Define Employment as a binary YES or NO variable where YES corresponds to "Employed" and NO corresponds to "Not Employed."
  - A subject will be considered "employed" at a given visit if Q1 = YES or Q2 > 0 or Q4 > 0.
  - A subject will be considered "unemployed" at a given visit if Q1 = NO and no positive hours recorded under Q2 and Q4 (i.e., if Q1 = NO AND Q2  $\leq$  0 AND Q4  $\leq$  0, then UNEMPLOYED).
  - Employment status for a subject will be considered "missing" at a given visit if Q1 = missing and no positive hours recorded under Q2 and Q4.

- If a subject is "unemployed" or employment status is "missing," then S1, S2, and S3 will be set to "missing."
- If Q2 = 0 and Q4 = 0 or missing then Q2/(Q2 + Q4) = missing (i.e., S1 = missing).
- If Q2 = 0 and Q4 = 0, then set S3 to missing.
- If Q2 is missing or Q4 is missing, then set S1 and S3 to missing.
- If Q4 = missing, then DO NOT set Q5 = missing.
- If Q5 is missing, then apply the following rules:
  - $\circ$  If Q2 > 0, Q4 = 0, and Q5 = missing, then S3 = 100%.
  - If Q2 = 0, Q4 > 0, and Q5 = missing, then S3 is missing.
  - $\circ$  If Q2 > 0, Q4 > 0, and Q5 = missing, then S3 is missing.
- Determine if a subject missed work (based on Q2) in order to analyze the proportion of subjects who missed work:
  - Create a binary (yes or no) "missed work" variable.
  - A subject will be considered as yes to missed work if Q2 is greater than 0.
  - If Q2 = missing, then MISSED WORK = missing.
  - $\circ$  If Q2 > 0, then MISSED WORK = "yes."
  - $\circ$  If Q2 = 0, then MISSED WORK = "no."

Therefore, the proportion of subjects who missed work will be counted based on the number of subjects with MISSED WORK = YES.

### 9.4.24 Health Resource Utilization (HRU) Questionnaire

The HRU questionnaire contains three questions regarding health care utilization in the following categories: unscheduled health care professional visits, emergency room visits, and hospital admissions. The data gathered from the HRU questionnaire will be used to calculate the individual cumulative number of utilizations per unit of time (e.g., subject-year) under observation in each variable (i.e., the number of unscheduled PsA-related health care professional visits, the number of emergency room visits, the number of hospital admissions and the total number of days in hospital) as follows:



- Time under observation for a subject will be defined as "date of last visit with non-missing HRU date of baseline visit."
- The number of utilizations after baseline will be summed up for each subject.

To determine cumulative HRU over all subjects, the ratio of the total number of utilizations (i.e., over all subjects) and the total time under observation (i.e., over all subjects) will be calculated across all subjects in each treatment group. HRU will be analyzed as observed only.

## 10.0 Safety Analysis

#### 10.1 General Considerations

Safety analyses will be carried out using the Safety Analysis Set by "as treated" treatment groups. There are two sets of planned safety analysis: safety analysis through Week 24, and long-term safety analysis.

#### **Safety Analysis Through Week 24**

Standard safety analyses by the "as treated" treatment groups of upadacitinib 15 mg QD, upadacitinib 30 mg QD, and the combined placebo group will be performed on safety data up to Week 24. No protocol-defined treatment switching will occur prior to this time point.

The standard safety analyses will include reporting of adverse events (AEs), laboratory, and vital signs measurements. Frequency tables of subjects with treatment-emergent adverse events (TEAEs) by system organ class (SOC) and by preferred term (PT) as in the Medical Dictionary for Regulatory Activities (MedDRA) dictionary will be provided by treatment groups. All continuous laboratory parameters and vital signs variables at each visit will be summarized by treatment groups. Frequency tables of subjects meeting criteria for potentially clinically significant vital sign values and for potentially clinically significant laboratory values will be provided by treatment groups. Missing safety data will not be imputed. Treatment comparations of upadacitinib versus placebo will be



provided for key safety endpoints including overview of AE, overview of AE of special interest, change from baseline in selected laboratory parameters and potentially clinically significant laboratory values. Treatment difference and corresponding 95% CI will be provided.

#### **Long-Term Safety Analysis**

Long-term safety analyses that account for protocol-defined treatment switching include reporting of AE rate adjusted by cumulative exposure, descriptive summary in laboratory parameters and vital sign variables by visit, and rate of potentially clinically significant laboratory and vital signs values. The treatment-emergent adverse event (TEAE) rate per 100 patient-years of exposure will be presented by actual treatment received at the time of AE (as described in Section 10.2.2). Listing of subjects with TEAEs by SOC and PT will be provided. Summary statistics for laboratory parameters and vital signs variables at each visit will be presented by "as treated" treatment group sequences defined below. Frequency tables and listings of subjects meeting criteria for potentially clinically significant vital sign values and for potentially clinically significant laboratory values will be provided by actual treatment received at the time of event. Missing safety data will not be imputed.

"As treated" treatment group sequences are defined as follows:

- 1. Placebo → Upadacitinib 15 mg QD
- 2. Placebo → Upadacitinib 30 mg QD
- 3. Upadacitinib 15 mg QD
- 4. Upadacitinib 30 mg QD

Starting with Amendment 7.01.01 (for Japan) and Amendment 8 and 8.01 (for global), subjects receiving upadacitinib 30 mg QD will be switched to upadacitinib 15 mg QD. For these subjects, adverse events and exposure to upadacitinib 30 mg QD will be



censored at the time of dose switch; subsequent adverse events and exposure starting the day of first dose of upadacitinib 15 mg QD will be summarized under separate groups, as described in Section 8.1.

Assessment of potentially clinically significant laboratory and vital sign values will be based on the same treatment groups as for adverse events. The baseline value for PCS determination will be the last non-missing value collected before the first dose of UPA (regardless of dose).

For descriptive summary by visit or mean change from baseline in laboratory values and vital signs, exposure sequences 2 and 4 (i.e., subjects who switched from upadacitinib 30 mg QD to 15 mg QD) will be censored at the time of dose switch. Descriptive summary by visit or mean change from baseline for laboratory values and vital signs collected after dose switch will be summarized separately by visits post switch. Note for analysis of mean change from baseline in laboratory values, the study baseline is used.

### 10.2 Analysis of Adverse Events

A treatment-emergent Adverse Event (TEAE) is defined as an adverse event with an onset date that is after the first dose of study drug, and no more than 30 days after the last dose of study drug.

Events where the onset date is the same as the study drug start date are assumed to be treatment-emergent, unless the study drug start time and the adverse event start time are collected and the adverse event start time is prior to the study drug start time. If an incomplete onset date was collected for an adverse event, the event will be assumed to be treatment-emergent unless there is other evidence that confirms that the event was not treatment-emergent (e.g., the event end date was prior to the study drug start date).

Adverse event data will be presented by SOCs and PTs using MedDRA Version 19.1 or most up to date version, which will be sorted in alphabetical order by SOC and PT.



# 10.2.1 Analysis of Adverse Events Prior to Protocol-Defined Treatment Switching

#### 10.2.1.1 Adverse Events Overview

The number and percentage of subjects experiencing TEAEs will be summarized by treatment groups for the following AE categories.

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs with a reasonable possibility of being related to study drug
- TEAEs leading to discontinuation of study drug
- TEAE leading to death
- Deaths (includes all deaths treatment-emergent and non-treatment-emergent)

In the AE overview summary, any event with an unknown severity will be considered as severe and any AE with an unknown relationship will be considered as having "reasonable possibility" of being related to study drug. Additional AE summaries may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

## 10.2.1.2 Adverse Events by System Organ Class and Preferred Term

The number and percentage of subjects experiencing adverse events will be tabulated by SOC and PT by treatment groups. The SOCs will be presented in alphabetical order, and the PTs will be presented in alphabetical order within each SOC.

The following summaries of adverse events will be generated:

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs with a reasonable possibility of being related to study drug



- TEAEs leading to discontinuation of study drug
- TEAE leading to death

Subjects reporting more than one adverse event for a given PT will be counted only once for that term (most severe incident for the severity tables and most related incident for the relationship tables). Subjects reporting more than one type of adverse event within a SOC will be counted only once for that SOC. Subjects reporting more than one type of adverse event will be counted only once in the overall total.

### 10.2.1.3 TEAEs by Maximum Severity

TEAEs will also be summarized by maximum severity by treatment groups. If a subject has an AE with an unknown severity, then the subject will be counted in the severity category of unknown, even if the subject has another occurrence of the same event with a severity present. The only exception is if the subject has another occurrence of the same AE with the highest CTCAE grade; in this case, the subject will be counted under the highest CTCAE grade for the term in question.

#### 10.2.1.4 TEAEs by Relationship

TEAEs will also be summarized by relationship to upadacitinib and placebo, as assessed by the investigator, by treatment groups. If a subject has a TEAE with an unknown relationship, then the subject will be counted in the relationship category of "unknown," even if the subject has another occurrence of the same event with a relationship present. The only exception is if the subject has another occurrence of the same TEAE with a relationship assessment of "reasonable possibility." In this case, the subject will be counted under the "reasonable possibility" category.

# 10.2.1.5 Frequent (≥ 2%) Adverse Events and Reasonably Possibly Related Adverse Events by System Organ Class and Preferred Term

TEAEs and reasonably possibly related AEs occurring for more than 2% of the subjects in any of the treatment groups will be summarized by SOC and PT separately.



### 10.2.1.6 Adverse Events of Special Interest

The Adverse Events of Special Interest (AESI) categories will be summarized and presented by treatment groups in overview as well as using SOC and PT. The AESI categories will be identified by the following search criteria per Standard MedDRA Queries (SMQs)/Company MedDRA Queries (CMQs) in Table 9 below. Adjudicated cardiovascular events will be summarized and presented by treatment group using the CAC adjudicated categories.



Table 9. AESI for Upadacitinib with SMQs/CMQs/PTs Searches

| AESI | Type of<br>MedDRA Query | Broad or<br>Narrow<br>Search | SMQ/CMQ Search<br>Criteria |
|---|---|---|---|
| Serious Infections | CMQ | | "Infections" – Subset for<br>SAEs |
| Opportunistic Infection excluding<br>Tuberculosis and Herpes Zoster | CMQ | | "Opportunistic Infection" |
| Possible Malignancy | SMQ | Narrow | "Malignancies" |
| Malignancy | SMQ | Narrow | "Malignant tumours" |
| Non-Melanoma Skin Cancer (NMSC) | SMQ | Narrow | Skin Malignant tumours<br>(Narrow SMQ) removing<br>Melanoma CMQ |
| Malignancy excluding NMSC | | | "Malignant tumours" SMQ<br>(Narrow) removing NMSC<br>output |
| Lymphoma | SMQ | Broad | "Malignant Lymphomas" |
| Hepatic Disorder | SMQ | Narrow | "Drug Related Hepatic<br>Disorders" |
| Adjudicated Gastrointestinal Perforations | Based on<br>adjudicated results<br>(the identification<br>of events to be<br>adjudicated are<br>described in the<br>GI Perforation<br>charter) | | |
| Anemia | CMQ | | "Non-Hemolytic and Non-<br>Aplastic Anemias" |
| Neutropenia | CMQ | | "Hematological Toxicity –<br>Neutropenia" |
| Lymphopenia | CMQ | | "Hematological Toxicity –<br>Lymphopenia" |
| Herpes Zoster | CMQ | | "Herpes Zoster" |
| Creatine Phosphokinase (CPK)<br>Elevation | PT | | Search only for the PT of "Blood creatine phosphokinase increased" |



**Table 9.** AESI for Upadacitinib with SMQs/CMQs/PTs Searches (Continued)

| AESI | Type of<br>MedDRA Query | Broad or<br>Narrow<br>Search | SMQ/CMQ Search<br>Criteria |
|---|---|---|---|
| Renal Dysfunction | SMQ | Narrow | "Acute Renal Failure" |
| Active Tuberculosis | CMQ | | "Active Tuberculosis" |
| Adjudicated Cardiovascular Events | Output from CAC | | |
| MACE* | | | |
| Cardiovascular Death | | | |
| Non-fatal Myocardial Infarction | | | |
| Non-fatal Stroke | | | |
| Other Adjudicated Cardiovascular Events | | | |
| Undetermined/Unknown Cause of Deaths | | | |
| Adjudicated Thrombotic Events | Output from CAC | | |
| VTE** | | | |
| Deep Vein Thrombosis | | | |
| Pulmonary Embolism | | | |
| Other Venous Thrombosis | | | |
| Arterial Thromboembolic Events (non-cardiac, non-neurologic) | | | |

CAC = Cardiovascular Adjudication Committee; CMQ = company MedDRA query; PT = preferred term; SMQ = standard MedDRA query

Additional AEs may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

<sup>\*</sup> MACE; Major Adverse Cardiovascular Events, defined as cardiovascular death, non-fatal myocardial infarction and non-fatal stroke.

<sup>\*\*</sup> VTE: Venous thromboembolic events, defined as deep vein thrombosis (DVT) and pulmonary embolism (PE) (fatal and non-fatal).



#### 10.2.2 Analysis of Long-Term Adverse Event Rates

Long-term adverse event rates will be analyzed using event rates adjusted by cumulative exposure and will be based on the actual treatment received at the time of AE occurrence. For subjects switched from upadacitinib 30 mg QD to upadacitinib 15 mg QD, adverse events and exposure to upadacitinib 30 mg QD will be censored at the time of dose switch; subsequent adverse events and exposure starting the day of first dose of upadacitinib 15 mg QD will be summarized under separate groups. The detailed treatment groups, including the handling of dose switch, are described in Section 8.1.

#### **Exposure-Adjusted Event Rate (EAER)**

To adjust for potentially different follow-up time between treatment groups, EAER will be provided. For the purpose of event rate calculation, the numerator will be the total number of AEs reported for the event (i.e., a subject can contribute more than one event to the numerator) and the denominator will be the total exposure time among subjects under the treatment group. The number of AEs reported (numerator), the total number of years of study drug exposure (denominator), and the exposure-adjusted AE event rate per 100 patient-years calculated as ([numerator/denominator]) • 100 will be presented for each treatment group. The EAER will be the main approach to evaluate AEs in the long-term analysis.

The exposure adjusted incidence rate (censored at the time of first event) may be conducted for selected AESI endpoints as appropriate for long-term analysis.

# 10.2.2.1 Overview of Adverse Events Rates per 100 Patient-Years of Study Drug Exposure

An overview of AEs per 100 patient-years of study exposure will be presented by treatment group for the following AE categories.

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events



- TEAEs with a reasonable possibility of being related to study drug
- TEAEs leading to discontinuation of study drug
- TEAE leading to death
- Deaths (includes all deaths treatment-emergent and non-treatment-emergent)

In the AE overview summary, any event with an unknown severity will be considered as severe and any AE with an unknown relationship will be considered as having "reasonable possibility" of being related to study drug. Additional AE categories may be considered for tabulation/summary based on recommendations from Clinical and Safety as deemed appropriate.

# 10.2.2.2 Adverse Events Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT

For each treatment group, the TEAE rate per 100 patient-years of exposure will be calculated overall, for each SOC and each PT, for each of the following AE categories:

- All TEAEs
- Treatment-emergent serious adverse events (SAEs)
- Treatment-emergent severe adverse events
- TEAEs with a reasonable possibility of being related to study drug
- TEAEs leading to discontinuation of study drug
- TEAE leading to death

# 10.2.2.3 Adverse Events of Special Interest Rates per 100 Patient-Years of Study Drug Exposure by SOC and PT

The Adverse Events of Special Interest (AESI) categories will be summarized and presented for each treatment group in overview as well as using SOC and MedDRA PT, for each of the AESI listed in Section 10.2.1.6. The AESI categories will be identified per Standard MedDRA Queries (SMQs)/Company MedDRA Queries (CMQs). Adjudicated



cardiovascular events will be summarized and presented by treatment group using the CAC adjudicated categories.

# 10.2.2.4 Listing of Serious Adverse Events (Including Deaths) and Adverse Events Leading to Study Drug Discontinuation

All serious adverse events (SAEs), deaths, and adverse events leading to discontinuation of study drug will be listed.

### 10.3 Analysis of Laboratory Data

#### 10.3.1 Variables and Units

All laboratory parameters to be collected in this study are listed below. Laboratory parameters will be reported using the standard international (SI) units.

Table 10. List of Laboratory Variables

| Laboratory Variables |
|----------------------------------|
| Hematology |
| White Blood Cell (WBC) Count |
| Red Blood Cell (RBC) Count |
| Hemoglobin |
| Hematocrit |
| Platelet count |
| Neutrophils |
| Basophils |
| Eosinophils |
| Lymphocytes |
| Monocytes |
| Bands |
| Chemistry |
| Total Bilirubin |
| Alkaline Phosphatase (ALP) |
| Aspartate aminotransferase (AST) |
| Alanine aminotransferase (ALT) |



# **Table 10.** List of Laboratory Variables (Continued)

| Laboratory Variables |
|-------------------------------------|
| Chemistry (Continued) |
| Total Protein |
| Albumin |
| Glucose |
| Triglycerides |
| Blood Urea Nitrogen (BUN) |
| Creatinine |
| Sodium |
| Potassium |
| Calcium |
| Inorganic Phosphorus |
| Creatine Phosphokinase (CPK) |
| Chloride |
| Bicarbonate |
| Cholesterol |
| LDL cholesterol |
| HDL cholesterol |
| LDL/HDL ratio |
| Cholesterol/HDL ratio |
| Urinalysis |
| Specific Gravity |
| pH |
| Protein |
| Glucose |
| Ketones |
| Blood |
| Microscopic Examination (if needed) |
| Urobilinogen |
| Bilirubin |
| Leukocytes |
| Nitrites |



#### **Table 10.** List of Laboratory Variables (Continued)

| Laboratory Variables |
|----------------------|
| Other |
| hs-CRP |
| ESR |

#### 10.3.2 Analysis of Laboratory Data Through Week 24

The laboratory data will be summarized by the treatment groups (upadacitinib 15 mg QD, upadacitinib 30 mg QD, and the combined placebo group).

#### 10.3.2.1 Assessment of Clinical Laboratory Variables

Analyses of hematology, chemistry, and urinalysis variables which are measured longitudinally will be performed by visits and by treatment groups. For analysis at each visit, the following summary statistics of visit values will be presented for each treatment group: sample size, mean, standard deviation, minimum, median, and maximum.

An ANOVA model with treatment as a factor will be used to compare change from baseline between different treatment groups for selected laboratory parameters. Mean difference from placebo and associated 95% CIs will be presented. The analysis applies to the following laboratory parameters of clinical interest: hemoglobin, platelets, lymphocytes, neutrophils, creatinine, ALT, AST, creatine phosphokinase (CPK), LDL, HDL, total cholesterol/HDL-cholesterol, LDL-cholesterol/HDL-cholesterol, and total cholesterol.

# 10.3.2.2 Assessment of Shift from Baseline in Clinical Laboratory Variables

The baseline and post-baseline laboratory observations will be categorized as Grade 0, Grade 1, Grade 2, Grade 3, and Grade 4 and shifts from baseline grade to worst ontherapy grade will be summarized. Toxicity grading scale is based on National Cancer



Institute Common Toxicity Criteria (NCI CTC) AE version 4.03. Shift tables from Baseline according to the grades will be provided for laboratory variables.

For LDL cholesterol, HDL cholesterol, total cholesterol, and triglycerides, the following categories according to National Cholesterol Education Program (NCEP) Adult Treatment Panel III (ATP III) guidelines will be used.

- LDL cholesterol ( $< 3.36, \ge 3.36 \text{ and } < 4.14, \ge 4.14 \text{ mmol/L}$ )
- HDL cholesterol ( $< 1.03, \ge 1.03 \text{ mmol/L}$ )
- Total cholesterol ( $< 5.17, \ge 5.17 \text{ and } < 6.21, \ge 6.21 \text{ mmol/L}$ )
- Triglycerides ( $< 1.69, \ge 1.69 \text{ and } < 2.26, \ge 2.26 \text{ mmol/L}$ )

Note that the minimum/maximum category is used, rather than the category of the minimum/maximum value. The two may be different due to variation in the reference range.

No statistical tests will be performed for this analysis.

# 10.3.2.3 Assessment of Potentially Clinical Significant Laboratory Values

The criteria for potentially clinically significant laboratory values will be determined by CTCAE criteria of Grade 2, Grade 3, Grade 4 and ≥ Grade 3 (if applicable), with a grade worsening compared to baseline. Toxicity grading scale is based on National Cancer Institute Common Toxicity Criteria (NCI CTC) AE version 4.03. The number and percentage of subjects meeting the criteria for potentially clinically significant laboratory values will be summarized by treatment groups.

#### 10.3.2.4 Assessment of Liver Elevations

According to FDA's Guidance for Industry "Drug-Induced Liver Injury: Premarketing clinical evaluation" (July 2009), when aminotransferase abnormalities indicating hepatocellular injury are accompanied by evidence of impaired hepatic function (bilirubin elevation > 2 × ULN), in the absence of evidence of biliary obstruction (i.e., significant
elevation of ALP) or some other explanation of the injury (e.g., viral hepatitis, alcohol hepatitis), the combined finding (i.e., Hy's Law cases) represents a signal of a potential for the drug to cause severe DILI.

For the purpose of assessing for potential Hy's law cases, the frequencies and percentages of subjects with post baseline liver specific function test values that meet the following criteria of potential clinical interest will be summarized by treatment groups:

- $ALT > 3 \times ULN$
- ALT  $\geq$  5 × ULN
- ALT  $\geq 10 \times ULN$
- ALT  $\geq 20 \times ULN$
- AST  $\geq$  3 × ULN
- AST  $\geq$  5 × ULN
- AST  $\geq 10 \times ULN$
- AST  $\geq 20 \times ULN$
- TBL  $\geq 2 \times ULN$
- Alkaline phosphatase  $\geq 1.5 \times ULN$
- ALT and/or AST  $\geq$  3 × ULN and concurrent TBL  $\geq$  1.5 × ULN
- ALT and/or AST  $\geq$  3 × ULN and concurrent TBL  $\geq$  2 × ULN

#### 10.3.3 Analysis of Long-Term Laboratory Data

#### 10.3.3.1 Assessment of Clinical Laboratory Variables

Analyses of hematology, chemistry, and urinalysis variables which are measured longitudinally will be performed by visits and by treatment group sequences as described in Section 10.1. For each analysis, the following summary statistics of visit values will be presented for each treatment group sequence: sample size, mean, standard deviation, minimum, median and maximum.



Analyses will be performed for change from baseline in hemoglobin, lymphocytes, neutrophils, creatinine, and creatine phosphokinase (CPK).

Descriptive summary by visit or mean change from baseline in laboratory values for subjects who switched from upadacitinib 30 mg QD to 15 mg QD will be censored at the time of dose switch, and descriptive summary by visit or mean change from baseline for values post switch will be summarized separately, as described in Section 10.1.

## 10.3.3.2 Assessment of Potentially Clinical Significant Laboratory Values

Long-term laboratory data will be summarized based on the number and percentage of subjects meeting the criteria for potentially clinical significant laboratory values and by the actual treatment received at the time of the event occurrence. The treatment groups for summarizing potentially clinically significant laboratory values are the same as the ones for long-term AE analysis as described in Section 10.1. A subject can be counted under different treatment groups if he/she was on placebo from baseline to Week 24 and then started upadacitinib 15 or 30 mg at Week 24 and experienced potentially clinical significant laboratory values under different treatment groups.

In the evaluation of potentially clinically significant laboratory values, the baseline value will be determined by the last non-missing measurement recorded on or before the date of the first dose of study drug in the corresponding treatment group (which may be different than the first dose of study drug received in the study). For example, for a subject who started on placebo and switched to upadacitinib 15 mg QD at Week 24, lab values under upadacitinib 15 mg QD exposure would be evaluated against the baseline value defined as the last non-missing measurement recorded on or before the date of the first dose of upadacitinib 15 mg QD. For subjects who switched from upadacitinib 30 mg QD to upadacitinib 15 mg QD, lab values under upadacitinib 15 mg QD exposure would still be evaluated against the baseline defined based on the first dose of upadacitinib 30 mg QD.



A listing of all subjects with any laboratory determination meeting CTCAE criteria of Grade 2 or above with a grade worsening compared to baseline will be provided. For each of these subjects, the whole course of the respective parameter will be listed.

#### 10.3.3.3 Assessment of Liver Elevations

The frequencies and percentages of subjects with post-baseline liver-specific function test values that meet the following criteria of potential clinical interest will be summarized by the actual treatment received at the time of the event occurrence. The treatment groups for summarizing liver elevations are the same as the ones for long-term AE analysis as described in Section 8.1.

A subject can be counted under different treatment groups if he/she was on placebo from baseline to Week 24 and then started upadacitinib 15 or 30 mg at Week 24 and experienced potentially clinical significant laboratory values under different treatment groups.

A listing of potentially clinically significant liver elevations based on criteria specified above will be provided. For each of these subjects, the whole course of the respective parameter will be listed.

#### 10.4 Analysis of Vital Signs

#### 10.4.1 Variables and Criteria Defining Abnormality

Vital sign variables include sitting systolic blood pressure, sitting diastolic blood pressure, pulse rate, and weight. The criteria for potentially clinically significant vital sign findings are presented in Table 11.



Table 11. Criteria for Potentially Clinically Significant Vital Sign Findings

| Vital Sign | Category | Criteria for Potential Clinically Significant Vital Signs |
|---|---|---|
| Systolic blood pressure | Low | Value ≤ 90 mmHg and decrease ≥ 20 mmHg from Baseline |
| | High | Value $\geq 160$ mmHg and increase $\geq 20$ mmHg from Baseline |
| Diastolic blood pressure | Low | Value ≤ 50 mmHg and decrease ≥ 10 mmHg from Baseline |
| | High | Value $\geq 100$ mmHg and increase $\geq 10$ mmHg from Baseline |
| Weight | High | > 7% increase from baseline |
| | Low | > 7% decrease from baseline |

#### 10.4.2 Analysis of Vital Signs Through Week 24

Analyses of vital sign variables which are measured longitudinally will be performed by visits and by the treatment groups of upadacitinib 15 mg QD, upadacitinib 30 mg QD, and the combined placebo group. For each analysis, the following summary statistics will be presented for each treatment group: sample size, mean, standard deviation, minimum, median, and maximum.

The number and percentage of subjects meeting the criteria for potentially clinically significant vital sign values will be summarized by treatment groups.

#### 10.4.3 Analysis of Long-Term Vital Signs

Analyses of vital signs variables which are measured longitudinally will be performed by visits and by treatment group sequences as described in Section 10.1. For each analysis, the following summary statistics will be presented for each treatment group: sample size, mean, standard deviation, minimum, median, and maximum.

Long-Term vital signs will also be summarized based on the number and percentage of subjects meeting the criteria for potentially clinical significant vital sign values and by the actual treatment received at the time of the event occurrence. The treatment groups are the same as the ones for long-term AE analysis as described in Section 10.2.2. A subject can be counted under different treatment groups if he/she was on placebo from baseline to Week 24 and then started upadacitinib 15 or 30 mg at Week 24 and experienced



potentially clinical significant laboratory values under different treatment groups. In the evaluation of potentially clinically significant vital sign values, the baseline value will be determined by the last non-missing measurement recorded on or before the date of the first dose of study drug in the corresponding treatment group, similarly as described in Section 10.3.3.2.

Descriptive summary by visit in vital signs for subjects who switched from upadacitinib 30 mg QD to 15 mg QD will be censored at the time of dose switch, and descriptive summary by visit for values post switch will be summarized separately, as described in Section 10.1.2. The treatment groups for summarizing PCS vital sign values are the same as the ones for long-term AE analysis as described in Section 8.1. For the purpose of evaluating PCS vital sign values, for subjects who switched from upadacitinib 30 mg QD to upadacitinib 15 mg QD, baseline is defined based on the first dose of Upadacitinib 30 mg QD, similarly as described in Section 10.3.3.2.

A listing of all subjects with any vital sign values meeting the criteria for potentially clinically significant vital signs will be provided. For each of these subjects, the whole course of the respective parameter will be listed.

## 11.0 Summary of Changes

# 11.1 Summary of Changes between the Previous Version and the Current Version

The primary efficacy analysis has been completed under the SAP version 2.0 and SPP version 1.0, Period 1 reporting has been completed under the SAP version 2.0 and SPP version 2.0. The current SAP update applies only to future reporting of long-term analysis.

1. Updated throughout the SAP to align with Protocol Amendment 7.01.01 and Amendment 8 and 8.01, including handling of dose switch from upadacitinib 30 mg QD to 15 mg QD (hereafter referred to as "dose switch").



- 1) Updated Section 7.0 and Section 8.1 to provide analysis details that incorporate dose switch.
- 2) Updated Section 9.1 to summarize the analysis changes that incorporate dose switch for long-term efficacy analysis.
- 3) Updated Section 10.1, Section 10.2.2, Section 10.3.3.1, Section 10.3.3.2, Section 10.3.3.3 and Section 10.4.3 to incorporate handling of dose switch for long-term safety analysis.
- 2. Updated Section 9.1.2 and Section 9.3 for long-term efficacy analysis.
  - 1) Updated Section 9.1.2 to describe the missing data handling approach for the additional long-term efficacy analysis using MMRM/GLMM models.
  - 2) Updated Section 9.3 to add NRI and/or GLMM for long-term binary endpoint analysis (Week 104 and future).
  - 3) Updated Section 9.3 to add MMRM based on AO data for long-term continuous endpoint analysis (Week 104 and future).
- 3. Updated language in Section 10.1, Section 10.2.1.1, Section 10.2.2.1, Section 10.2.2.3 to add clarity for safety analysis.
- 4. Updated Section 10.2.1.6 and Section 10.4.1 to align with the latest upadacitinib AESI definitions in PSSAP V4.0.
- 5. Added Appendix E to describe analysis accounting for impact of COVID-19 pandemic.

### 12.0 Version History

Table 12. SAP Version History Summary

| Version | Date | Summary |
|---|---|---|
| 2.0 | 02 Oct 2019 | Used for primary analysis |
| 3.0 | 24 May 2021 | Incorporating updates 1) in statistical analysis to handle the missing data due to COVID-19; 2) in wording changes in PSSAP. 3) in handling of dose switch from upadacitinib 30 mg QD to 15 mg QD. 4) Add additional long-term analysis method for Week 104 and future visits. |

### 13.0 References

- 1. Bretz F, Maurer W, Brannath W, et al. A graphical approach to sequentially rejective multiple test procedures. Stat Med. 2009;28(4):586-604.
- 2. Greenland S, Rothman KJ. Introduction to stratified analysis. In: Rothman KJ, Greeland S, Lash TL, editors. Modern Epidemiology, 3<sup>rd</sup> Edition. Philaphdelphia: Lippincott Williams & Wilkins; 2008.
- 3. Carpenter JR, Kenward MG. Multiple Imputation and Its Application. New York: John Wiley & Sons; 2013.
- 4. Ratitch B, Lipkovich O'Kelly M. Combining analysis results from multiply imputed categorical data. In: Conference Proceedings from PharmaSUG 2013. Paper SP03. May 12-5, 2013: Chicago, IL.
- 5. Liu GF, Wang J, Liu K, et al. Confidence intervals for an exposure adjusted incidence rate difference with application to clinical trials. Stat Med. 2006;25(8):1275-86.

#### **Appendix A.** SAS Procedure for Mantel-Haenszel Test

A SAS procedure, the Proc Freq, will be used to compute the statistics using the Mantel-Haenszel method.<sup>2</sup> Risk difference, 95% CI and p value will be provided through the program.

#### SAS code example:

```
title 'Placebo vs ABT-494 30 mg QD';
proc freq data= wk12_nri;
where TRTP='Placebo'|TRTP='ABT-494 30 mg QD';
table TRTP*aval/ nopercent nocol chisq riskdiff(cl=wald)
alpha=0.05;
run;

title2 'For p-values';
proc freq data=wk12_nri;
where TRTP='Placebo'|TRTP='ABT-494 30 mg QD';
tables DMARDBL*TRTP*aval/ cmh;
run;
```



#### Appendix B. Tipping Point Analysis for ACR20 at Week 12

To assess the robustness of the primary analysis using NRI data handling, tipping point analysis is conducted on the primary endpoint ACR20. The analysis is conducted on the FAS using As Observed data handling.

The tipping point analysis will be performed by multiple imputations using logistic regression, allowing the imputed ACR response rate to systematically vary from 0% to 100% in both upadacitinib and placebo, respectively. This will be accomplished by modifying the predicted probabilities for the responses through shifting the log odds ratios,<sup>3</sup> then directly sampling the missing ACR20 response from the Bernoulli distribution with the modified probabilities.

For each pair of shift parameters, the same CMH method used for the primary endpoint will be performed on each of the multiple imputed datasets to obtain the results for each comparison of the upadacitinib treatment group versus the placebo group. Because chi-square distribution of CMH test statistic is skewed from the normal distribution, to combine the results from the CMH test using Rubin's method, a transformation will be conducted to normalize the CMH statistic.<sup>4</sup> These transformed results will be then aggregated using Rubin's method to get *P*-values.

#### Appendix C. Tipping Point Analysis for Key Secondary Continuous Endpoint

To assess the impact of potential departures from the missing-at-random assumption, tipping point analyses are conducted as a sensitivity check for change from baseline in the key secondary continuous endpoint HAQ-DI.

The tipping point analyses are two-dimensional, i.e., assumptions about the missing outcomes on each upadacitinib dose group and the placebo group are allowed to vary independently. In addition, the focus is on scenarios where missing outcomes on upadacitinib are worse than the imputed values on upadacitinib, while missing outcomes on placebo are better than the imputed values on placebo. Missing values are first imputed via MI under MAR (where the MI imputation is performed upon AO data), and then a shift parameter is applied to the imputed values (a different shift parameter may be specified for each treatment group). This is implemented by PROC MI using the MNAR statement.

More specifically, PROC MI using the fully conditional specification (FCS) method will be performed to impute any missing value and therefore does not rely on a monotone missing pattern. In fact, the FCS method can handle any arbitrary missing data pattern. Treatment is included in the FCS imputation model to enable sampling conditional on treatment groups. Additionally, the imputation model includes stratification factor of current use of non-biologic DMARD (yes/no), gender, race (white vs. non-white), age, baseline BMI, geographic regions, duration of PsA diagnosis and the baseline value of the endpoints of interest, as well as longitudinal response observed at any other visits.

For a given pair of shift parameters, the SAS code example is as follows:

```
PROC MI DATA=DATA_WIDE OUT=DATA_WIDE_BOUNDED NIMPUTE=20
SEED=12345;

CLASS TRTP &COVCAT;
FCS;
By trtp;
VAR &COVCON &COVCAT WEEK_2 WEEK_4 WEEK_8 WEEK_12;
MNAR ADJUST (WEEK_12 / SHIFT=&SJ1
ADJUSTOBS=(TRTP='PLACEBO'));
```

```
MNAR ADJUST (WEEK_12 / SHIFT=&SJ2 ADJUSTOBS=(TRTP='UPA
15MG'));
RUN;
```

Note:

The input dataset is in wide format. TRTP denotes the treatment group. &COVCON denotes baseline continuous covariates including baseline age, baseline BMI, duration of PsA diagnosis and baseline value of the endpoint of interest. &COVCAT denotes categorical covariates including current use of non-biological DMARD gender, race, and regions. WEEK\_2, WEEK\_4, WEEK\_8, WEEK\_12 denote the observed values at each visit. &SJ1 and &SJ2 denote the shift parameters for the placebo group and upadacitinib 15 MG group respectively.

In cases where the shifted values are smaller than the minimum or larger than maximum value of the endpoint, (i.e., out of range), the minimum or maximum value of the endpoint is used in further analysis steps. For each pair of shift parameters, the SAS procedure PROC MIXED is used for ANCOVA model with Huber-White sandwich errors which includes the fixed effects of treatment, the stratification factor of current DMARD use and the continuous fixed covariate of baseline measurement on each of the multiple imputed datasets to obtain the results for each upadacitinib treatment group versus the placebo group comparison. These results will be aggregated using Rubin's method to get p-values.

If one pair of shift parameters are found to just reverse the study conclusion, in terms of p-value larger than 0.05 (the original p-value < 0.05), then the shift parameters are identified as the tipping point. The results for a grid of shift parameter combinations are provided in tabular format.

The SAS code example of the data imputation step for tipping point analysis using MI is provided above. The SAS code example for the analysis and results combination step using PROC MIXED and PROC MIANALYZE is as follows:

```
PROC MIXED DATA=ALL EMPIRICAL;

ODS OUTPUT LSMEANS=MIXEDLSMEANS DIFFS=DIFF;

BY Shift1 Shift2 _IMPUTATION_;

CLASS TRTP STRATA USUBJID;

MODEL CHG = BASELINE TRTP STRATA / SOLUTION;

LSMEANS TRTP / CL PDIFF DIFF;

REPEATED /SUBJECT=USUBJID;

RUN;
```

Note:

```
DATA DIFF1;
    SET DIFF;
    COMPARISON= TRTP||' VS '||LEFT( TRTP);
RUN:
PROC SORT DATA=DIFF1; BY COMPARISON Shift1 Shift2 IMPUTATION; RUN;
PROC MIANALYZE DATA=DIFF1;
    ODS OUTPUT PARAMETERESTIMATES=GROUP OUTPUT;
    BY comparison shift1 shift2;
    MODELEFFECTS ESTIMATE;
    STDERR STDERR;
RUN;
/* Comparison of "UPA 15 mg" vs. "Placebo" */
data miparm1;
set GROUP_OUTPUT;
if comparison='1
                            VS
                                           2' then output miparm1;
run;
proc transpose data=miparm1(keep= Shift1 Shift2 Probt)
out=wide miparm1;
by shift1;
id shift2;
var Probt;
run;
```

The input dataset ALL includes all (# of shift1 parameters) \* (# of shift2 parameters) \* (# of imputations in MI) imputed datasets. TRTP denotes the treatment group and STRATA denotes the stratification factor used in analysis. CHG denotes the change from baseline value and BASELINE denotes the baseline value.



# Appendix D. Exposure Adjusted AE Rate Difference and Normal Approximation Based 95% Confidence Interval (Liu, F et al. 2006<sup>5</sup>)

Assume the occurrence of TEAE of special interest follows a Poisson distribution and let  $\lambda$  denote the rate of occurrence of TEAE under the total exposure time for a treatment group. Let  $n_1$  and  $n_2$  be the number of AEs reported in an upadacitinib dose group and the combined placebo group, respectively. Let  $T_1$  and  $T_2$  be the total number of days exposed to study drug summed across all treated subjects in an upadacitinib dose group and the combined placebo group. Under the assumption that  $n_1$  and  $n_2$  follow independent Poisson distribution with parameters  $\lambda_1 T_1$  and  $\lambda_2 T_2$ , the  $\hat{\lambda}_1 = n_1/T_1$  and  $\hat{\lambda}_2 = n_2/T_2$ . So the exposure adjusted TEAE rate difference can be estimated by

$$\theta = \hat{\lambda}_1 - \hat{\lambda}_2$$

Using normal approximation, the 95% confidence interval can be calculated by

$$\hat{\lambda}_1 - \hat{\lambda}_2 \pm Z_{\alpha/2}\hat{\sigma}$$

where 
$$\hat{\sigma} = \sqrt{n_1/T_1^2 + n_2/T_2^2}$$



## Appendix E. Statistical Analysis to Account for the Impact of COVID-19 Pandemic

This section presents the changes in statistical analysis to handle the missing data due to COVID-19 and the additional data collected related to COVID-19. The Week 24 primary database lock was completed in Oct 2019. The analyses specified in this section only applies to analysis for the long-term database lock.

#### **Patient Disposition**

Reasons for premature discontinuation of study drug/study will be updated to add two additional reasons related to COVID-19.

- COVID-19 Infection
- COVID-19 Logistical restrictions

The number and percentage of subjects who prematurely discontinued from study drug/study due to COVID-19 infection or COVID-19 logistical restrictions will be summarized by randomized treatment group.

#### **Summary of COVID-19 Impacted Visits**

Types of missing visits related to COVID-19 will be collected for the protocol prespecified visits. For each visit, the number and percentage of subjects impacted by COVID-19 will be summarized by the types of visit for each randomized treatment group as well as overall:

- In person, partial assessments done
- Virtual visit
- Missed visit



#### **Efficacy Analyses**

With respect to COVID-19 pandemic, it would be reasonable to assume that missed visits and missing data due to self-quarantine or local government restrictions on travel or limitations on healthcare resources will impact subjects across treatment arms in a similar fashion and adopt the Missing at Random (MAR) assumption for missing data handling.

As described in Section 9.3, longitudinal analysis models MMRM and GLMM, as well as NRI analysis for binary variables will be used for long term efficacy analysis for the treatment sequences, and will be maintained for long term efficacy analysis in the presence of missing data due to COVID-19.

#### **Safety Analyses**

COVID-19 related AEs occurring on or after February 01, 2020 and COVID-19 related deaths occurring on or after February 01, 2020 will be collected.

Listings of subjects with COVID-19 related AEs and deaths will be provided.